CLINICAL TRIAL: NCT01777139
Title: A Multicentre, Open-label, Long-term, Safety, Tolerability, and Efficacy Study of Retigabine Immediate-release (IR) in Asian Adults With Partial Onset Seizures (Extension of Study RTG114855)
Brief Title: A Long-term, Safety, Tolerability, and Efficacy Study of Retigabine Immediate-release (IR) in Asian Adults With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114873
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Epilepsy
Keywords: Retigabine; Drug-Resistant; Epilepsy; Partial-Onset Seizures; Safety and Tolerability; Immediate Release; Long-Term; Adjunctive Therapy; Asian Subjects; Efficacy; GW582892
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retigabine IR (Experimental): All subjects will initially receive a starting dose of retigabine IR at 900 mg/day and after the first week of the OLE study, the dose of retigabine IR may be increased or decreased in increments or decrements of decrements of 150 mg/day on weekly basis based on efficacy and tolerability. The overall daily dose of retigabine IR must be maintained between a minimum dose of 600 mg/day and a maximum dose of 1200 mg/day.
  Interventions: Drug: Retigabine IR

INTERVENTIONS:
Drug: Retigabine IR — Retigabine IR tablets will be available in 5 strengths: 50 mg, 100 mg, 200 mg, 300 mg, and 400 mg.

SUMMARY:
This is a multicentre, long-term, open-label extension (OLE) study to assess the long-term safety, tolerability and efficacy of retigabine immediate-release (IR) as adjunctive therapy in adult Asian subjects with drug-resistant partial-onset seizures (POS).

DETAILED DESCRIPTION:
Subjects who successfully complete the Maintenance Phase of Study RTG114855 (parent study) and are expected to benefit from therapy with retigabine IR will be eligible for this OLE study. The study will consist of Screening (1 day), Open-Label Treatment and Follow-up (3 weeks) phase. Subjects will initially receive a starting dose of retigabine IR at 900 milligram (mg)/day and the same concurrent antiepileptic drug (AED) regimen that they were receiving at the final visit of the Transition Phase of the parent study. After the first week of the OLE study, the dose of retigabine IR may be adjusted to between 600 and 1200 mg/day, with dose adjustments in increments or decrements of 150 mg/week, based on efficacy and tolerability. In addition, the dose and number of concurrent AEDs may also be adjusted to meet each individual subject's needs. The efficacy and safety issues will be assessed throughout the study; subjects will be instructed to call the investigator if they experience any efficacy or tolerability issues between the study visits. As the duration of the study will be determined based on the following four conditions: 1) regulatory approval and commercialisation of retigabine IR; 2) retigabine IR is not approved by the regulatory authorities; 3) the study is terminated by the Sponsor for reasons including, but not limited to, safety issues; or 4) the subject is withdrawn or withdraws consent, 4 years will be considered as a guide to the duration of the study. The safety and tolerability endpoints are incidence and severity of adverse events (AEs); proportion of subjects with AEs leading to discontinuation; change from Baseline in vital sign measurements and weight; change from Baseline in electrocardiogram parameters; change from Baseline in haematology, chemistry, and urinalysis parameters; changes from Baseline in American Urological Association Symptom Index and post-void residual bladder ultrasound volumes; and summary of the Columbia-Suicide Severity Rating Scale. Efficacy will be assessed by calculating the percent change from Baseline (parent study) in 28-day total POS frequency for the entire open-label Treatment Phase of this OLE study. This will also be calculated based on duration of exposure. Responder rate (defined as a >/=50% reduction from Baseline in 28-day total POS frequency) will also be summarised for the entire open-label Treatment Phase and by duration of exposure.

ELIGIBILITY:
Inclusion Criteria:

* The subject has successfully completed the Maintenance Phase and Transition Phase of Study RTG114855.
* The subject is expected, in the opinion of the investigator, to benefit from participation in this OLE study.
* The subject or the caregiver is able and willing to maintain an accurate and complete written daily seizure calendar for the entire duration of the study.
* The subject has given written informed consent, or has a legally authorized representative who has given written informed consent, prior to the performance of any study assessments.
* A female subject is eligible to enrol and participate in the study if she is of: nonchildbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is premenarchal or postmenopausal), premenopausal females with a documented (medical report verification) hysterectomy with or without oophorectomy, or bilateral oophorectomy when reproductive status has been confirmed by hormone level assessment, and postmenopausal females defined as being amenorrhoeic for >1 year with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms). However, if indicated, this should be confirmed by oestradiol and follicle stimulating hormone levels consistent with menopause (according to local laboratory ranges). Women who have not been confirmed as postmenopausal should be advised to use contraception.
* Childbearing potential, has a negative urine or serum pregnancy test at Screening.
* Is not pregnant or lactating or planning to become pregnant during the study.

Exclusion Criteria:

* Has met any of the withdrawal criteria in the parent study (RTG114855) or has, in the opinion of the investigator, clinically significant abnormal laboratory or ECG findings that preclude entry into RTG114873.
* Is planning to begin treatment with an investigational drug (other than retigabine) and/or an experimental device for the treatment of epilepsy or any other medical condition.
* Has any medical condition that, in the investigator's judgement, is considered to be clinically significant and could potentially affect subject safety or study outcome, including but not limited to clinically significant cardiac, renal, or hepatic condition; or a condition that affects the absorption, distribution, metabolism, or excretion of drugs.
* Is unwilling or unable to follow the study procedures or reporting of AEs.
* Has active suicidal plan/intent or has had active suicidal thoughts in the past 6 months or has history of suicide attempt in the last 2 years or >1 lifetime suicide attempt.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- GSK Investigational Site, Kuala Lumpur, Malaysia
- South Korea (5):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with partial-onset seizures (POS) who successfully completed the maintenance phase of study RTG114855 (NCT01648101) were recruited in this open-label extension (OLE) study.
Pre-assignment Details: All the participants received at least 1 dose of retigabine (RTG) immediate release (IR). Screening was performed on the day of final visit of the parent study. A total of 30 participants, 12 from placebo and 18 from RTG group who completed the treatment and transition phases of the parent study were included in this OLE study.
Groups:
- RTG IR: Eligible participants initially received a starting dose of RTG IR 900 milligrams per day (mg/day) and the same doses of the same concurrent anti-epileptic drugs (AEDs) that they were receiving at the final visit of the transition phase of the parent study. After the first week of the OLE study, the dose of RTG IR could be increased or decreased in increments or decrements 150 mg/day on weekly basis based on efficacy and tolerability. The overall daily dose of RTG IR was to be maintained between a minimum dose of 600 mg/day and a maximum dose of 1200 mg/day.
- RTG in Safety Follow-up Continuation Phase (SFUCP): Participants who withdraw from the Open-Label Treatment Phase and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP which was the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR.
Period: Primary Reporting Phase (Up to 4 Years)
Arm/Group | RTG IR | RTG in Safety Follow-up Continuation Phase (SFUCP)
Started | 30 | 0
Completed | 0 | 0
Not Completed | 30 | 0
Not completed — Adverse Event | 7 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Withdrawal by Subject | 8 | 0
Not completed — Other (Study drug discontinued) | 3 | 0
Not completed — Other (Reached stopping criteria) | 2 | 0
Not completed — Other (Subjects entered SFUCP) | 4 | 0
Period: SFUCP (Up to 1.4 Years)
Arm/Group | RTG IR | RTG in Safety Follow-up Continuation Phase (SFUCP)
Started | 0 | 4
Completed | 0 | 0
Not Completed | 0 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other-Study drug discontinued | 0 | 3

BASELINE CHARACTERISTICS:
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.0 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 17
  Asian-South East Asian Heritage | 12
  Asian-Mixed Race | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent (TE) Serious Adverse Events (SAEs) and Non-SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function is SAE. TEAE refers to an AE for which the onset was on or after the date of the first RTG dose in this study and on or before 30 days after the last RTG dose date. AEs that started in the parent study that worsened in this study were also considered as TEAEs. Safety population comprised of participants who take at least 1 dose of study medication after they have enrolled into this OLE study. Number of participants with TE-SAEs and non-SAEs (with incidence >= 5%) have been presented.
Time Frame: Up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  Any non-SAE | 23
  Any SAE | 5

2. Primary Outcome: Percentage of Participants With TEAEs Leading to Study Discontinuation
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE refers to an AE for which the onset was on or after the date of the first RTG dose in this study and on or before 30 days after the last RTG dose date. Percentage of participants with TEAEs leading to study discontinuation were presented.
Time Frame: Up to 4 years
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Percentage of Participants | 17

3. Primary Outcome: Number of Participants With Potential Clinical Concern (PCC) Values of Change From Baseline for Vital Signs
Description: The vital signs were evaluated as per PCC Criteria. The vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR). The vital signs were measured in a seated position after 5 minutes of rest. PCC range for DBP was increase or decrease of >=20, for SBP was increase or decrease of >=15 and for heart rate was increase or decrease of >=15. A Baseline assessment in this OLE study was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Number of participants with vital sign values of PCC at any Post-Baseline visit were presented.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  DBP; increase by >=20 | 4
  DBP; decrease by >=20 | 9
  SBP; increase by >=15 | 5
  SBP; decrease by >=15 | 5
  HR; increase by >=15 | 9
  HR; decrease by >=15 | 5

4. Primary Outcome: Number of Participants With PCC Values of Change From Baseline for Body Weight
Description: Body weight of participants were measured as a measure of safety. PCC range for body weight was increase or decrease of >=7 percent. A Baseline assessment in this OLE study was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Number of participants with PCC values of body weight at any Post-Baseline visit were presented.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  Body weight;increase by >=7 percent | 11
  Body weight; decrease by >=7 percent | 4

5. Primary Outcome: Number of Participants With PCC Values of Change From Baseline for Electrocardiogram (ECG) Parameters
Description: Single measurements of 12-lead ECGs were obtained in a supine position after at least 10 minutes of rest using an ECG machine that automatically calculates the heart rate (HR) as beats per minute (bpm) and measures PR, QRS, Bazett's correction QT interval (QTcB) and Friedericia's correction QT interval (QTcF) in milliseconds (msec). A Baseline assessment in this OLE study was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Number of participants with PCC values of ECG parameters at any Post-Baseline visit were presented. For the 'Any Post Baseline' value, only the worst case finding was counted for each participant.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  HR <50 bpm, decreased from Baseline>=15 bpm | 1
  HR >100 bpm, increased from Baseline >=15 bpm | 0
  PR interval >=210 msec, increased from Baseline | 1
  QRS interval >=120 msec, increased from Baseline | 0
  QTcB:Post-Baseline QTc>=450, Baseline<450 msec | 5
  QTcB:Post-Baseline QTc>=480, Baseline < 480 msec | 0
  QTcB:Post-Baseline QTc>500 msec | 0
  QTcB:Post-Baseline QTc>=500, Baseline <500msec | 0
  QTcB:Increase in QTc of >30 msec from Baseline | 3
  QTcB:Increase in QTc of >30,<=60 msecfrom Baseline | 3
  QTcB:Increase in QTc of >60 msec from Baseline | 0
  QTcF:Post-Baseline QTc>=450, Baseline<450 msec | 1
  QTcF:Post-Baseline QTc>=480, Baseline<480 msec | 0
  QTcF: Post-Baseline QTc>500 msec | 0
  QTcF:Post-Baseline QTc>=500, Baseline<500 msec | 0
  QTcF:Increase in QTc of >30 msec from Baseline | 3
  QTcF:Increase in QTcof >30,<=60 msec from Baseline | 3
  QTcF:Increase in QTc of >60 msec from Baseline | 0

6. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Total Neutrophils, and White Blood Cell Count (WBC)
Description: Blood samples were collected from participants for evaluation of change from Baseline in hematology parameters including basophils, eosinophils, lymphocytes,monocytes, platelet count, total neutrophils, and WBC. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and standard deviation (SD) were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga unit per liter (GI/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Giga unit per liter (GI/L)
  Basophils;Visit 1-Day 1;n=29: number analyzed (Participants) | 29
  Basophils;Visit 1-Day 1;n=29 | 0.000 (0.0118)
  Basophils;Visit 2 - Month 1;n=28: number analyzed (Participants) | 28
  Basophils;Visit 2 - Month 1;n=28 | 0.000 (0.0126)
  Basophils;Visit 3 - Month 3;n=26: number analyzed (Participants) | 26
  Basophils;Visit 3 - Month 3;n=26 | 0.000 (0.0118)
  Basophils;Visit 4 - Month 6;n=16: number analyzed (Participants) | 16
  Basophils;Visit 4 - Month 6;n=16 | -0.003 (0.0184)
  Basophils;Visit 5 - Month 9;n=16: number analyzed (Participants) | 16
  Basophils;Visit 5 - Month 9;n=16 | 0.001 (0.0178)
  Basophils;Visit 6 - Month 12;n=13: number analyzed (Participants) | 13
  Basophils;Visit 6 - Month 12;n=13 | 0.003 (0.0132)
  Basophils;Visit 7 (Month 16);n=12: number analyzed (Participants) | 12
  Basophils;Visit 7 (Month 16);n=12 | -0.002 (0.0147)
  Basophils;Visit 8 (Month 20);n=11: number analyzed (Participants) | 11
  Basophils;Visit 8 (Month 20);n=11 | 0.003 (0.0220)
  Basophils;Visit 9 (Month 24);n=10: number analyzed (Participants) | 10
  Basophils;Visit 9 (Month 24);n=10 | 0.000 (0.0105)
  Basophils;Visit 10 (Month 28);n=10: number analyzed (Participants) | 10
  Basophils;Visit 10 (Month 28);n=10 | 0.002 (0.0079)
  Basophils;Visit 11 (Month 32);n=9: number analyzed (Participants) | 9
  Basophils;Visit 11 (Month 32);n=9 | 0.004 (0.0188)
  Basophils;Visit 12 (Month 36);n=4: number analyzed (Participants) | 4
  Basophils;Visit 12 (Month 36);n=4 | 0.005 (0.0058)
  Basophils;Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Basophils;Study Conclusion/Withdrawal;n=28 | -0.003 (0.0146)
  Basophils;Follow-Up Visit;n=5: number analyzed (Participants) | 5
  Basophils;Follow-Up Visit;n=5 | -0.008 (0.0130)
  Eosinophils;Visit 1-Day 1; n=29: number analyzed (Participants) | 29
  Eosinophils;Visit 1-Day 1; n=29 | -0.012 (0.1152)
  Eosinophils; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Eosinophils; Visit 2 - Month 1; n=28 | -0.051 (0.1311)
  Eosinophils; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Eosinophils; Visit 3 - Month 3; n=26 | -0.070 (0.2813)
  Eosinophils; Visit 4 - Month 6; n=16: number analyzed (Participants) | 16
  Eosinophils; Visit 4 - Month 6; n=16 | -0.004 (0.1020)
  Eosinophils; Visit 5 - Month 9; n=16: number analyzed (Participants) | 16
  Eosinophils; Visit 5 - Month 9; n=16 | 0.038 (0.1038)
  Eosinophils; Visit 6 - Month 12; n=13: number analyzed (Participants) | 13
  Eosinophils; Visit 6 - Month 12; n=13 | -0.014 (0.0846)
  Eosinophils; Visit 7 (Month 16); n=12: number analyzed (Participants) | 12
  Eosinophils; Visit 7 (Month 16); n=12 | 0.010 (0.1135)
  Eosinophils; Visit 8 (Month 20); n=11: number analyzed (Participants) | 11
  Eosinophils; Visit 8 (Month 20); n=11 | 0.008 (0.0908)
  Eosinophils; Visit 9 (Month 24); n=10: number analyzed (Participants) | 10
  Eosinophils; Visit 9 (Month 24); n=10 | -0.051 (0.0983)
  Eosinophils; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Eosinophils; Visit 10 (Month 28); n=10 | 0.006 (0.1467)
  Eosinophils; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Eosinophils; Visit 11 (Month 32); n=9 | 0.011 (0.0494)
  Eosinophils; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Eosinophils; Visit 12 (Month 36); n=4 | -0.025 (0.0900)
  Eosinophils; Study Conclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  Eosinophils; Study Conclusion/Withdrawal; n=28 | -0.026 (0.1085)
  Eosinophils; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Eosinophils; Follow-Up Visit; n=5 | -0.078 (0.1268)
  Lymphocytes; Visit 1-Day 1; n= 29: number analyzed (Participants) | 29
  Lymphocytes; Visit 1-Day 1; n= 29 | -0.132 (0.5985)
  Lymphocytes; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Lymphocytes; Visit 2 - Month 1; n=28 | -0.065 (0.5549)
  Lymphocytes; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Lymphocytes; Visit 3 - Month 3; n=26 | -0.120 (0.4974)
  Lymphocytes; Visit 4 - Month 6; n=16: number analyzed (Participants) | 16
  Lymphocytes; Visit 4 - Month 6; n=16 | 0.024 (0.3740)
  Lymphocytes; Visit 5 - Month 9; n=16: number analyzed (Participants) | 16
  Lymphocytes; Visit 5 - Month 9; n=16 | -0.032 (0.4358)
  Lymphocytes; Visit 6 - Month 12; n= 13: number analyzed (Participants) | 13
  Lymphocytes; Visit 6 - Month 12; n= 13 | -0.109 (0.3685)
  Lymphocytes; Visit 7 (Month 16); n=12: number analyzed (Participants) | 12
  Lymphocytes; Visit 7 (Month 16); n=12 | 0.007 (0.3039)
  Lymphocytes; Visit 8 (Month 20); n=11: number analyzed (Participants) | 11
  Lymphocytes; Visit 8 (Month 20); n=11 | -0.037 (0.3250)
  Lymphocytes; Visit 9 (Month 24); n=10: number analyzed (Participants) | 10
  Lymphocytes; Visit 9 (Month 24); n=10 | 0.052 (0.4157)
  Lymphocytes; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Lymphocytes; Visit 10 (Month 28); n=10 | 0.108 (0.2986)
  Lymphocytes; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Lymphocytes; Visit 11 (Month 32); n=9 | 0.022 (0.4280)
  Lymphocytes; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Lymphocytes; Visit 12 (Month 36); n=4 | -0.268 (0.3096)
  Lymphocytes; Study Conclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  Lymphocytes; Study Conclusion/Withdrawal; n=28 | -0.068 (0.5778)
  Lymphocytes; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Lymphocytes; Follow-Up Visit; n=5 | -0.070 (0.3466)
  Monocytes; Visit 1-Day 1; n= 29: number analyzed (Participants) | 29
  Monocytes; Visit 1-Day 1; n= 29 | -0.018 (0.1204)
  Monocytes; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Monocytes; Visit 2 - Month 1; n=28 | -0.028 (0.1357)
  Monocytes; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Monocytes; Visit 3 - Month 3; n=26 | -0.044 (0.1350)
  Monocytes; Visit 4 - Month 6; n=16: number analyzed (Participants) | 16
  Monocytes; Visit 4 - Month 6; n=16 | 0.033 (0.1445)
  Monocytes; Visit 5 - Month 9; n=16: number analyzed (Participants) | 16
  Monocytes; Visit 5 - Month 9; n=16 | -0.042 (0.1348)
  Monocytes; Visit 6 - Month 12; n= 13: number analyzed (Participants) | 13
  Monocytes; Visit 6 - Month 12; n= 13 | 0.076 (0.1711)
  Monocytes; Visit 7 (Month 16); n=12: number analyzed (Participants) | 12
  Monocytes; Visit 7 (Month 16); n=12 | -0.021 (0.1717)
  Monocytes; Visit 8 (Month 20); n=11: number analyzed (Participants) | 11
  Monocytes; Visit 8 (Month 20); n=11 | 0.129 (0.1936)
  Monocytes; Visit 9 (Month 24); n=10: number analyzed (Participants) | 10
  Monocytes; Visit 9 (Month 24); n=10 | -0.021 (0.1358)
  Monocytes; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Monocytes; Visit 10 (Month 28); n=10 | -0.022 (0.1781)
  Monocytes; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Monocytes; Visit 11 (Month 32); n=9 | 0.088 (0.1384)
  Monocytes; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Monocytes; Visit 12 (Month 36); n=4 | 0.035 (0.0823)
  Monocytes; Study Conclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  Monocytes; Study Conclusion/Withdrawal; n=28 | 0.014 (0.1809)
  Monocytes; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Monocytes; Follow-Up Visit; n=5 | 0.054 (0.1011)
  Platelet count; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Platelet count; Visit 1-Day 1; n=28 | 8.3 (25.26)
  Platelet count; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Platelet count; Visit 2 - Month 1; n=28 | 6.3 (24.01)
  Platelet count; Visit 3 - Month 3; n=25: number analyzed (Participants) | 25
  Platelet count; Visit 3 - Month 3; n=25 | 14.5 (26.01)
  Platelet count; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Platelet count; Visit 4 - Month 6; n=18 | 5.8 (37.84)
  Platelet count; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Platelet count; Visit 5 - Month 9; n=17 | 6.0 (29.90)
  Platelet count; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Platelet count; Visit 6 - Month 12; n=15 | 10.2 (35.51)
  Platelet count; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  Platelet count; Visit 7 (Month 16); n=14 | 18.5 (23.65)
  Platelet count; Visit 8 (Month 20); n=11: number analyzed (Participants) | 11
  Platelet count; Visit 8 (Month 20); n=11 | 16.6 (39.64)
  Platelet count; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  Platelet count; Visit 9 (Month 24); n=11 | 15.5 (22.98)
  Platelet count; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Platelet count; Visit 10 (Month 28); n=10 | 20.3 (40.66)
  Platelet count; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Platelet count; Visit 11 (Month 32); n=9 | 17.1 (50.38)
  Platelet count; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Platelet count; Visit 12 (Month 36); n=4 | 28.5 (13.53)
  Platelet count; Study Conclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  Platelet count; Study Conclusion/Withdrawal; n=28 | 17.0 (37.37)
  Platelet count; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Platelet count; Follow-Up Visit; n=5 | -2.0 (26.93)
  Total Neutrophils; Visit 1-Day 1; n=30 | -0.099 (1.3450)
  Total Neutrophils; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Total Neutrophils; Visit 2 - Month 1; n=28 | -0.028 (1.1045)
  Total Neutrophils; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Total Neutrophils; Visit 3 - Month 3; n=26 | 0.369 (1.7061)
  Total Neutrophils; Visit 4 - Month 6; n=16: number analyzed (Participants) | 16
  Total Neutrophils; Visit 4 - Month 6; n=16 | -0.318 (1.4286)
  Total Neutrophils; Visit 5 - Month 9; n=16: number analyzed (Participants) | 16
  Total Neutrophils; Visit 5 - Month 9; n=16 | -0.158 (1.6801)
  Total Neutrophils; Visit 6 - Month 12; n=13: number analyzed (Participants) | 13
  Total Neutrophils; Visit 6 - Month 12; n=13 | 0.182 (0.9911)
  Total Neutrophils; Visit 7 (Month 16); n=12: number analyzed (Participants) | 12
  Total Neutrophils; Visit 7 (Month 16); n=12 | 0.252 (0.9079)
  Total Neutrophils; Visit 8 (Month 20); n=11: number analyzed (Participants) | 11
  Total Neutrophils; Visit 8 (Month 20); n=11 | 0.325 (1.0561)
  Total Neutrophils; Visit 9 (Month 24); n=10: number analyzed (Participants) | 10
  Total Neutrophils; Visit 9 (Month 24); n=10 | 0.656 (1.0269)
  Total Neutrophils; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Total Neutrophils; Visit 10 (Month 28); n=10 | 0.238 (0.8603)
  Total Neutrophils; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Total Neutrophils; Visit 11 (Month 32); n=9 | 1.310 (2.2464)
  Total Neutrophils; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Total Neutrophils; Visit 12 (Month 36); n=4 | 0.310 (0.6800)
  Total Neutrophils;Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Total Neutrophils;Study Conclusion/Withdrawal;n=28 | 0.086 (1.1378)
  Total Neutrophils; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Total Neutrophils; Follow-Up Visit; n=5 | -0.176 (1.4051)
  WBC ; Visit 1-Day 1; n=30 | -0.15 (1.417)
  WBC ; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  WBC ; Visit 2 - Month 1; n=28 | -0.16 (1.182)
  WBC; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  WBC; Visit 3 - Month 3; n=26 | 0.14 (1.501)
  WBC; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  WBC; Visit 4 - Month 6; n=18 | -0.42 (1.545)
  WBC; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  WBC; Visit 5 - Month 9; n=17 | -0.12 (1.630)
  WBC; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  WBC; Visit 6 - Month 12; n=15 | 0.34 (1.330)
  WBC ; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  WBC ; Visit 7 (Month 16); n=14 | 0.20 (0.927)
  WBC ; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  WBC ; Visit 8 (Month 20); n=12 | 0.53 (1.127)
  WBC ; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  WBC ; Visit 9 (Month 24); n=11 | 0.64 (0.837)
  WBC; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  WBC; Visit 10 (Month 28); n=10 | 0.33 (1.003)
  WBC; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  WBC; Visit 11 (Month 32); n=9 | 1.43 (2.155)
  WBC; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  WBC; Visit 12 (Month 36); n=4 | 0.08 (0.991)
  WBC; Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  WBC; Study Conclusion/Withdrawal;n=28 | 0.01 (1.212)
  WBC; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  WBC; Follow-Up Visit; n=5 | -0.28 (1.395)

7. Primary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected from participants for evaluation of hematocrit. Hematocrit is a ratio of red blood cells to the total volume of blood. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Proportion of red blood cells in blood
  Visit 1-Day 1; n=30 | -0.0035 (0.02749)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | -0.0048 (0.02512)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | -0.0033 (0.02175)
  Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Visit 4 - Month 6; n=18 | -0.0022 (0.01659)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | -0.0004 (0.01790)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | -0.0014 (0.01883)
  Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  Visit 7 (Month 16); n=14 | 0.0027 (0.01887)
  Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 (Month 20); n=12 | 0.0105 (0.01857)
  Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 (Month 24); n=11 | 0.0174 (0.02331)
  Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Visit 10 (Month 28); n=10 | 0.0189 (0.01987)
  Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Visit 11 (Month 32); n=9 | 0.0344 (0.02959)
  Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Visit 12 (Month 36); n=4 | 0.0408 (0.02608)
  Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Study Conclusion/Withdrawal;n=28 | 0.0055 (0.02345)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 0.0048 (0.02100)

8. Primary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected from participants to evaluate change from Baseline in hemoglobin and MCHC levels. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per Liter (G/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Gram per Liter (G/L)
  Hemoglobin; Visit 1-Day 1; n=30 | -2.6 (8.23)
  Hemoglobin; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Hemoglobin; Visit 2 - Month 1; n=28 | -2.8 (7.75)
  Hemoglobin; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Hemoglobin; Visit 3 - Month 3; n=26 | -2.2 (6.83)
  Hemoglobin; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Hemoglobin; Visit 4 - Month 6; n=18 | -0.2 (5.33)
  Hemoglobin; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Hemoglobin; Visit 5 - Month 9; n=17 | -0.8 (5.96)
  Hemoglobin; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Hemoglobin; Visit 6 - Month 12; n=15 | -1.9 (6.28)
  Hemoglobin; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  Hemoglobin; Visit 7 (Month 16); n=14 | -1.5 (6.00)
  Hemoglobin; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  Hemoglobin; Visit 8 (Month 20); n=12 | 2.3 (5.10)
  Hemoglobin; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  Hemoglobin; Visit 9 (Month 24); n=11 | 2.6 (6.55)
  Hemoglobin; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Hemoglobin; Visit 10 (Month 28); n=10 | 1.9 (6.12)
  Hemoglobin; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Hemoglobin; Visit 11 (Month 32); n=9 | 9.1 (9.84)
  Hemoglobin; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Hemoglobin; Visit 12 (Month 36); n=4 | 8.0 (6.98)
  Hemoglobin; Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Hemoglobin; Study Conclusion/Withdrawal;n=28 | 1.3 (6.31)
  Hemoglobin; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Hemoglobin; Follow-Up Visit; n=5 | 1.8 (7.92)
  MCHC; Visit 1-Day 1; n=30 | -3.1 (8.45)
  MCHC; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  MCHC; Visit 2 - Month 1; n=28 | -2.9 (7.92)
  MCHC; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  MCHC; Visit 3 - Month 3; n=26 | -2.4 (9.27)
  MCHC; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  MCHC; Visit 4 - Month 6; n=18 | 1.2 (7.31)
  MCHC; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  MCHC; Visit 5 - Month 9; n=17 | -1.1 (4.61)
  MCHC; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  MCHC; Visit 6 - Month 12; n=15 | -2.6 (7.21)
  MCHC; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  MCHC; Visit 7 (Month 16); n=14 | -5.1 (9.63)
  MCHC; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  MCHC; Visit 8 (Month 20); n=12 | -2.3 (7.80)
  MCHC; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  MCHC; Visit 9 (Month 24); n=11 | -6.4 (8.56)
  MCHC; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  MCHC; Visit 10 (Month 28); n=10 | -9.9 (8.24)
  MCHC; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  MCHC; Visit 11 (Month 32); n=9 | -4.6 (6.31)
  MCHC; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  MCHC; Visit 12 (Month 36); n=4 | -12.8 (4.19)
  MCHC; StudyConclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  MCHC; StudyConclusion/Withdrawal;n=28 | -1.3 (8.47)
  MCHC; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  MCHC; Follow-Up Visit; n=5 | 0.8 (10.43)

9. Primary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH) Level
Description: Blood samples were collected from participants to evaluate change from Baseline in MCH levels. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram (Pg)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Picogram (Pg)
  Visit 1-Day 1; n=30 | -0.30 (0.539)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | -0.16 (0.807)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | -0.23 (0.759)
  Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Visit 4 - Month 6; n=18 | -0.14 (0.731)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | -0.46 (0.600)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | -0.65 (0.588)
  Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  Visit 7 (Month 16); n=14 | -0.56 (0.717)
  Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 (Month 20); n=12 | -0.73 (0.574)
  Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 (Month 24); n=11 | -0.87 (0.461)
  Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Visit 10 (Month 28); n=10 | -0.76 (0.435)
  Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Visit 11 (Month 32); n=9 | -0.73 (0.391)
  Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Visit 12 (Month 36); n=4 | -1.53 (0.506)
  StudyConclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  StudyConclusion/Withdrawal; n=28 | -0.52 (0.731)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | -0.64 (0.611)

10. Primary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV) and Mean Platelet Volume (MPV)
Description: Blood samples were collected from participants to evaluate change from Baseline in MCV and MPV levels. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Femtoliter (fL)
  MCV; Visit 1-Day 1; n=30 | 0.1 (2.15)
  MCV; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  MCV; Visit 2 - Month 1; n=28 | 0.4 (2.35)
  MCV; Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  MCV; Visit 3 - Month 3; n=26 | 0.1 (2.42)
  MCV; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  MCV; Visit 4 - Month 6; n=18 | -0.7 (1.75)
  MCV; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  MCV; Visit 5 - Month 9; n=17 | -1.1 (1.52)
  MCV; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  MCV; Visit 6 - Month 12; n=15 | -1.2 (2.08)
  MCV; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  MCV; Visit 7-(Month 16); n=14 | -0.1 (2.06)
  MCV; Visit 8-(Month 20); n=12: number analyzed (Participants) | 12
  MCV; Visit 8-(Month 20); n=12 | -1.3 (2.01)
  MCV; Visit 9-(Month 24); n=11: number analyzed (Participants) | 11
  MCV; Visit 9-(Month 24); n=11 | -0.7 (1.85)
  MCV; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  MCV; Visit 10-(Month 28); n=10 | 0.8 (2.44)
  MCV; Visit 1- (Month 32); n=9: number analyzed (Participants) | 9
  MCV; Visit 1- (Month 32); n=9 | -0.8 (2.05)
  MCV; Visit 12- (Month 36); n=4: number analyzed (Participants) | 4
  MCV; Visit 12- (Month 36); n=4 | -0.8 (1.26)
  MCV; StudyConclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  MCV; StudyConclusion/Withdrawal; n=28 | -1.0 (2.16)
  MCV; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  MCV; Follow-Up Visit; n=5 | -2.2 (1.64)
  MPV; Visit 1- Day 1; n=28: number analyzed (Participants) | 28
  MPV; Visit 1- Day 1; n=28 | -0.43 (0.526)
  MPV; Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  MPV; Visit 2 - Month 1; n=28 | -0.41 (0.610)
  MPV; Visit 3 - Month 3; n=25: number analyzed (Participants) | 25
  MPV; Visit 3 - Month 3; n=25 | -0.34 (0.579)
  MPV; Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  MPV; Visit 4 - Month 6; n=18 | -0.07 (0.642)
  MPV; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  MPV; Visit 5 - Month 9; n=17 | -0.32 (0.645)
  MPV; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  MPV; Visit 6 - Month 12; n=15 | -0.19 (0.678)
  MPV; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  MPV; Visit 7-(Month 16); n=14 | -0.36 (0.624)
  MPV; Visit 8-(Month 20); n=11: number analyzed (Participants) | 11
  MPV; Visit 8-(Month 20); n=11 | -0.15 (0.658)
  MPV; Visit 9-(Month 24); n=11: number analyzed (Participants) | 11
  MPV; Visit 9-(Month 24); n=11 | 0.07 (0.629)
  MPV; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  MPV; Visit 10-(Month 28); n=10 | -0.14 (0.435)
  MPV; Visit 11- (Month 32); n=9: number analyzed (Participants) | 9
  MPV; Visit 11- (Month 32); n=9 | 0.21 (0.933)
  MPV; Visit 12- (Month 36); n=4: number analyzed (Participants) | 4
  MPV; Visit 12- (Month 36); n=4 | -0.73 (0.386)
  MPV; StudyConclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  MPV; StudyConclusion/Withdrawal; n=28 | -0.18 (0.572)
  MPV; Follow-Up Visit; n=5: number analyzed (Participants) | 5
  MPV; Follow-Up Visit; n=5 | 0.28 (0.349)

11. Primary Outcome: Change From Baseline in Red Blood Cell (RBC) Count
Description: Blood samples were collected from participants to evaluate change from Baseline in RBC count. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Tetra unit per liter (TI/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Tetra unit per liter (TI/L)
  Visit 1- Day 1; n=30 | -0.03 (0.266)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | -0.06 (0.256)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | -0.03 (0.241)
  Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Visit 4 - Month 6; n=18 | 0.01 (0.227)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | 0.05 (0.218)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 0.04 (0.188)
  Visit 7 - (Month 16); n=14: number analyzed (Participants) | 14
  Visit 7 - (Month 16); n=14 | 0.04 (0.198)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | 0.19 (0.207)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | 0.22 (0.214)
  Visit 10 -(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10 -(Month 28); n=10 | 0.17 (0.200)
  Visit 11- (Month 32); n=9: number analyzed (Participants) | 9
  Visit 11- (Month 32); n=9 | 0.41 (0.322)
  Visit 12- (Month 36); n=4: number analyzed (Participants) | 4
  Visit 12- (Month 36); n=4 | 0.45 (0.265)
  StudyConclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  StudyConclusion/Withdrawal; n=28 | 0.13 (0.229)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 0.16 (0.241)

12. Primary Outcome: Change From Baseline in Red Cell Distribution Width (RDW)
Description: Blood samples were collected from participants to evaluate change from Baseline in RDW. RDW is a parameter that measures variation in red blood cell size or red blood cell volume. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Percentage of width
  Visit 1- Day 1; n=30 | 0.31 (0.887)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | 0.43 (0.716)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | 0.18 (1.016)
  Visit 4 - Month 6; n=18: number analyzed (Participants) | 18
  Visit 4 - Month 6; n=18 | -0.33 (0.806)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | -0.03 (1.025)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 0.01 (0.684)
  Visit 7 - (Month 16); n=14: number analyzed (Participants) | 14
  Visit 7 - (Month 16); n=14 | 0.13 (0.685)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | -0.33 (0.735)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | -0.01 (0.468)
  Visit 10 -(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10 -(Month 28); n=10 | 0.35 (0.665)
  Visit 11- (Month 32); n=9: number analyzed (Participants) | 9
  Visit 11- (Month 32); n=9 | -0.36 (0.814)
  Visit 12- (Month 36); n=4: number analyzed (Participants) | 4
  Visit 12- (Month 36); n=4 | -0.33 (0.690)
  Study Conclusion/Withdrawal; n=28: number analyzed (Participants) | 28
  Study Conclusion/Withdrawal; n=28 | -0.01 (1.009)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | -0.14 (0.885)

13. Primary Outcome: Change From Baseline in Alanine Amino Transferase (ALT), Alkaline Phosphatase (Alk. Phosph.), Aspartate Aminotransferase (AST), Creatine Kinase (CK), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LD)
Description: Blood samples collected from participants to evaluate change from Baseline in clinical chemistry parameters included ALT, Alk. phosph., AST,CK, GGT and LD. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
International unit per liter (IU/L)
  ALT; Visit 1-Day 1; n= 28: number analyzed (Participants) | 28
  ALT; Visit 1-Day 1; n= 28 | 0.8 (4.78)
  ALT; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  ALT; Visit 2 - Month 1; n=27 | 3.3 (14.86)
  ALT; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  ALT; Visit 3 - Month 3; n=24 | 0.3 (5.44)
  ALT; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  ALT; Visit 4 - Month 6; n=19 | 0.9 (6.20)
  ALT; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  ALT; Visit 5 - Month 9; n=17 | 0.6 (4.17)
  ALT; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  ALT; Visit 6 - Month 12; n=15 | 1.5 (6.41)
  ALT; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  ALT; Visit 7 (Month 16); n=14 | 0.3 (4.61)
  ALT; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  ALT; Visit 8 (Month 20); n=12 | 0.4 (4.62)
  ALT; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  ALT; Visit 9 (Month 24); n=11 | 0.8 (8.59)
  ALT; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  ALT; Visit 10 (Month 28); n=10 | 1.6 (6.00)
  ALT; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  ALT; Visit 11 (Month 32); n=9 | 7.4 (13.57)
  ALT; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  ALT; Visit 12 (Month 36); n=4 | 0.0 (5.29)
  ALT; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  ALT; Study Conclusion/Withdrawal; n=27 | 1.1 (6.05)
  ALT ; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  ALT ; Follow-Up Visit; n=4 | 9.8 (15.65)
  Alk. Phosph.; Visit 1-Day 1; n= 28: number analyzed (Participants) | 28
  Alk. Phosph.; Visit 1-Day 1; n= 28 | -1.5 (13.64)
  Alk. Phosph; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Alk. Phosph; Visit 2 - Month 1; n=27 | -2.2 (12.43)
  Alk. Phosph; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Alk. Phosph; Visit 3 - Month 3; n=24 | -2.5 (17.09)
  Alk. Phosph; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Alk. Phosph; Visit 4 - Month 6; n=19 | -5.1 (13.82)
  Alk. Phosph; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Alk. Phosph; Visit 5 - Month 9; n=17 | -4.7 (14.50)
  Alk. Phosph; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Alk. Phosph; Visit 6 - Month 12; n=15 | -2.5 (18.28)
  Alk. Phosph; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  Alk. Phosph; Visit 7 (Month 16); n=14 | 0.2 (20.10)
  Alk. Phosph; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  Alk. Phosph; Visit 8 (Month 20); n=12 | 0.5 (19.15)
  Alk. Phosph; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  Alk. Phosph; Visit 9 (Month 24); n=11 | -3.5 (16.42)
  Alk. Phosph; Visit 10 (Month 28); n=10: number analyzed (Participants) | 10
  Alk. Phosph; Visit 10 (Month 28); n=10 | -5.3 (12.68)
  Alk. Phosph; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  Alk. Phosph; Visit 11 (Month 32); n=9 | 5.8 (15.91)
  Alk. Phosph; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  Alk. Phosph; Visit 12 (Month 36); n=4 | 7.8 (18.03)
  Alk. Phosph; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  Alk. Phosph; Study Conclusion/Withdrawal; n=27 | -2.7 (16.65)
  Alk. Phosph ; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Alk. Phosph ; Follow-Up Visit; n=4 | -21.3 (19.69)
  AST; Visit 1-Day 1; n= 27: number analyzed (Participants) | 27
  AST; Visit 1-Day 1; n= 27 | 0.5 (6.35)
  AST; Visit 2 - Month 1; n=26: number analyzed (Participants) | 26
  AST; Visit 2 - Month 1; n=26 | 2.0 (10.61)
  AST; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  AST; Visit 3 - Month 3; n=24 | 0.0 (4.57)
  AST; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  AST; Visit 4 - Month 6; n=19 | 1.3 (4.13)
  AST; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  AST; Visit 5 - Month 9; n=17 | 2.6 (6.02)
  AST; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  AST; Visit 6 - Month 12; n=15 | 2.1 (5.42)
  AST; Visit 7 (Month 16); n=14: number analyzed (Participants) | 14
  AST; Visit 7 (Month 16); n=14 | 1.8 (3.17)
  AST; Visit 8 (Month 20); n=12: number analyzed (Participants) | 12
  AST; Visit 8 (Month 20); n=12 | 1.6 (3.32)
  AST; Visit 9 (Month 24); n=11: number analyzed (Participants) | 11
  AST; Visit 9 (Month 24); n=11 | 2.5 (4.30)
  AST; Visit 10 (Month 28); n=9: number analyzed (Participants) | 9
  AST; Visit 10 (Month 28); n=9 | 2.9 (4.88)
  AST; Visit 11 (Month 32); n=9: number analyzed (Participants) | 9
  AST; Visit 11 (Month 32); n=9 | 4.7 (4.58)
  AST; Visit 12 (Month 36); n=4: number analyzed (Participants) | 4
  AST; Visit 12 (Month 36); n=4 | 0.8 (2.50)
  AST; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  AST; Study Conclusion/Withdrawal; n=27 | 1.5 (6.08)
  AST; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  AST; Follow-Up Visit; n=4 | 7.5 (10.34)
  CK; Visit 1-Day 1; n= 28: number analyzed (Participants) | 28
  CK; Visit 1-Day 1; n= 28 | -103.3 (483.91)
  CK; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  CK; Visit 2 - Month 1; n=27 | -72.5 (414.16)
  CK; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  CK; Visit 3 - Month 3; n=24 | -88.8 (461.41)
  CK; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  CK; Visit 4 - Month 6; n=19 | -10.3 (56.38)
  CK; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  CK; Visit 5 - Month 9; n=17 | -10.9 (63.16)
  CK; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  CK; Visit 6 - Month 12; n=15 | 11.9 (62.40)
  CK; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  CK; Visit 7-(Month 16); n=14 | 9.2 (23.66)
  CK; Visit 8 -(Month 20); n=12: number analyzed (Participants) | 12
  CK; Visit 8 -(Month 20); n=12 | 1.3 (21.83)
  CK; Visit 9 -(Month 24); n=11: number analyzed (Participants) | 11
  CK; Visit 9 -(Month 24); n=11 | 4.8 (35.02)
  CK; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  CK; Visit 10-(Month 28); n=10 | 2.6 (27.47)
  CK; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  CK; Visit 11-(Month 32); n=9 | 93.7 (185.31)
  CK; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  CK; Visit 12-(Month 36); n=4 | 26.3 (51.06)
  CK; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  CK; Study Conclusion/Withdrawal; n=27 | 24.7 (658.19)
  CK; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  CK; Follow-Up Visit; n=4 | 261.0 (553.52)
  GGT; Visit 1-Day 1; n= 28: number analyzed (Participants) | 28
  GGT; Visit 1-Day 1; n= 28 | 4.6 (21.15)
  GGT; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  GGT; Visit 2 - Month 1; n=27 | 4.2 (37.01)
  GGT; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  GGT; Visit 3 - Month 3; n=24 | -4.5 (24.84)
  GGT; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  GGT; Visit 4 - Month 6; n=19 | -2.7 (18.93)
  GGT; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  GGT; Visit 5 - Month 9; n=17 | -2.5 (31.07)
  GGT; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  GGT; Visit 6 - Month 12; n=15 | -4.7 (21.26)
  GGT; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  GGT; Visit 7-(Month 16); n=14 | -3.6 (20.89)
  GGT; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  GGT; Visit 8 - (Month 20); n=12 | -13.1 (29.03)
  GGT; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  GGT; Visit 9 - (Month 24); n=11 | -6.0 (29.25)
  GGT; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  GGT; Visit 10-(Month 28); n=10 | 8.3 (23.32)
  GGT; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  GGT; Visit 11-(Month 32); n=9 | 24.3 (32.31)
  GGT; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  GGT; Visit 12-(Month 36); n=4 | 10.0 (27.48)
  GGT; StudyConclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  GGT; StudyConclusion/Withdrawal; n=27 | 2.1 (33.39)
  GGT; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  GGT; Follow-Up Visit; n=4 | -3.8 (9.03)
  LD; Visit 1-Day 1; n=27: number analyzed (Participants) | 27
  LD; Visit 1-Day 1; n=27 | -1.4 (20.13)
  LD; Visit 2 - Month 1; n=26: number analyzed (Participants) | 26
  LD; Visit 2 - Month 1; n=26 | 0.8 (22.57)
  LD; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  LD; Visit 3 - Month 3; n=24 | 1.7 (17.96)
  LD; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  LD; Visit 4 - Month 6; n=19 | -8.5 (19.35)
  LD; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  LD; Visit 5 - Month 9; n=17 | 1.9 (17.71)
  LD; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  LD; Visit 6 - Month 12; n=15 | -1.6 (22.21)
  LD; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  LD; Visit 7-(Month 16); n=14 | 1.3 (21.21)
  LD; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  LD; Visit 8 - (Month 20); n=12 | -0.5 (12.08)
  LD; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  LD; Visit 9 - (Month 24); n=11 | 12.2 (8.40)
  LD; Visit 10-(Month 28); n=9: number analyzed (Participants) | 9
  LD; Visit 10-(Month 28); n=9 | 8.3 (16.65)
  LD; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  LD; Visit 11-(Month 32); n=9 | 18.8 (18.98)
  LD; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  LD; Visit 12-(Month 36); n=4 | 8.5 (7.90)
  LD; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  LD; Study Conclusion/Withdrawal; n=27 | 2.6 (23.41)
  LD; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  LD; Follow-Up Visit; n=4 | 2.5 (8.19)

14. Primary Outcome: Change From Baseline in Albumin and Total Protein
Description: Blood samples were collected from participants to evaluate change from Baseline in albumin and total protein. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | RTG IR
Number analyzed (Participants) | 30
G/L
  Albumin; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Albumin; Visit 1-Day 1; n=28 | -0.9 (2.03)
  Albumin; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Albumin; Visit 2 - Month 1; n=27 | -0.3 (2.22)
  Albumin; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Albumin; Visit 3 - Month 3; n=24 | -0.3 (1.85)
  Albumin; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Albumin; Visit 4 - Month 6; n=19 | 0.1 (2.41)
  Albumin; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Albumin; Visit 5 - Month 9; n=17 | -0.3 (2.34)
  Albumin; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Albumin; Visit 6 - Month 12; n=15 | -1.1 (3.02)
  Albumin; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Albumin; Visit 7-(Month 16); n=14 | -0.7 (2.97)
  Albumin; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Albumin; Visit 8 - (Month 20); n=12 | -0.6 (2.02)
  Albumin; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Albumin; Visit 9 - (Month 24); n=11 | -0.3 (2.33)
  Albumin; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Albumin; Visit 10-(Month 28); n=10 | -0.2 (2.66)
  Albumin; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Albumin; Visit 11-(Month 32); n=9 | 1.2 (3.77)
  Albumin; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Albumin; Visit 12-(Month 36); n=4 | -0.3 (0.96)
  Albumin; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  Albumin; Study Conclusion/Withdrawal; n=27 | -0.6 (2.48)
  Albumin; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Albumin; Follow-Up Visit; n=4 | -0.3 (2.87)
  Total protein; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Total protein; Visit 1-Day 1; n=28 | -0.7 (2.84)
  Total protein; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Total protein; Visit 2 - Month 1; n=27 | -0.7 (4.08)
  Total protein; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Total protein; Visit 3 - Month 3; n=24 | 0.1 (3.35)
  Total protein; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Total protein; Visit 4 - Month 6; n=19 | 0.5 (3.66)
  Total protein; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Total protein; Visit 5 - Month 9; n=17 | -0.4 (3.87)
  Total protein; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Total protein; Visit 6 - Month 12; n=15 | -0.3 (5.23)
  Total protein; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Total protein; Visit 7-(Month 16); n=14 | 0.6 (5.36)
  Total protein; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Total protein; Visit 8 - (Month 20); n=12 | 1.3 (4.41)
  Total protein; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Total protein; Visit 9 - (Month 24); n=11 | 2.4 (4.37)
  Total protein; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Total protein; Visit 10-(Month 28); n=10 | 2.5 (4.86)
  Total protein; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Total protein; Visit 11-(Month 32); n=9 | 3.8 (6.63)
  Total protein; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Total protein; Visit 12-(Month 36); n=4 | 1.8 (2.22)
  Total protein; Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  Total protein; Study Conclusion/Withdrawal; n=27 | 0.7 (3.52)
  Total protein; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Total protein; Follow-Up Visit; n=4 | 0.5 (3.00)

15. Primary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN)/Creatinine Ratio
Description: Blood samples were collected from participants to evaluate change from Baseline in BUN/creatinine. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Ratio
  Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Visit 1-Day 1; n=28 | 4.2 (21.83)
  Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Visit 2 - Month 1; n=27 | 6.2 (20.92)
  Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Visit 3 - Month 3; n=24 | 7.0 (22.03)
  Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Visit 4 - Month 6; n=19 | 7.0 (18.11)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | 18.11 (16.40)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 5.5 (13.43)
  Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Visit 7-(Month 16); n=14 | 4.2 (24.49)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | 12.8 (21.46)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | 7.0 (16.25)
  Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10-(Month 28); n=10 | 1.9 (21.97)
  Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Visit 11-(Month 32); n=9 | 13.8 (25.29)
  Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Visit 12-(Month 36); n=4 | 30.0 (24.04)
  Study Conclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  Study Conclusion/Withdrawal; n=27 | 3.1 (24.50)
  Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Follow-Up Visit; n=4 | 1.0 (29.39)

16. Primary Outcome: Change From Baseline in Calcium, Carbon Dioxide (CO2) Content/Bicarbonate (Bicarb), Chloride, Glucose, Magnesium, Potassium, Sodium, Urea/BUN
Description: Blood samples were collected from participants to evaluate change from Baseline in calcium, CO2 content/Bicarb, chloride, glucose, magnesium, potassium, sodium, and urea/BUN. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Millimoles per liter (mmol/L)
  Calcium; Visit 1-Day 1; n=27: number analyzed (Participants) | 27
  Calcium; Visit 1-Day 1; n=27 | -0.015 (0.0759)
  Calcium; Visit 2 - Month 1; n=26: number analyzed (Participants) | 26
  Calcium; Visit 2 - Month 1; n=26 | -0.009 (0.0813)
  Calcium; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Calcium; Visit 3 - Month 3; n=24 | 0.017 (0.0586)
  Calcium; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Calcium; Visit 4 - Month 6; n=19 | 0.009 (0.0819)
  Calcium; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Calcium; Visit 5 - Month 9; n=17 | 0.020 (0.0742)
  Calcium; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Calcium; Visit 6 - Month 12; n=15 | -0.013 (0.0786)
  Calcium; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Calcium; Visit 7-(Month 16); n=14 | 0.009 (0.0809)
  Calcium; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Calcium; Visit 8 - (Month 20); n=12 | 0.013 (0.0628)
  Calcium; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Calcium; Visit 9 - (Month 24); n=11 | 0.006 (0.0543)
  Calcium; Visit 10-(Month 28); n=9: number analyzed (Participants) | 9
  Calcium; Visit 10-(Month 28); n=9 | 0.012 (0.0602)
  Calcium; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Calcium; Visit 11-(Month 32); n=9 | 0.026 (0.0915)
  Calcium; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Calcium; Visit 12-(Month 36); n=4 | 0.013 (0.0171)
  Calcium; StudyConclusion/Withdrawal; n=27: number analyzed (Participants) | 27
  Calcium; StudyConclusion/Withdrawal; n=27 | 0.015 (0.0820)
  Calcium; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Calcium; Follow-Up Visit; n=4 | 0.068 (0.0634)
  CO2 content/Bicarb; Visit 1-Day 1; n=27: number analyzed (Participants) | 27
  CO2 content/Bicarb; Visit 1-Day 1; n=27 | -0.3 (2.11)
  CO2 content/Bicarb; Visit 2 - Month 1; n=26: number analyzed (Participants) | 26
  CO2 content/Bicarb; Visit 2 - Month 1; n=26 | -0.3 (2.94)
  CO2 content/Bicarb; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  CO2 content/Bicarb; Visit 3 - Month 3; n=24 | -0.3 (3.52)
  CO2 content/Bicarb; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  CO2 content/Bicarb; Visit 4 - Month 6; n=19 | -0.6 (2.80)
  CO2 content/Bicarb; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  CO2 content/Bicarb; Visit 5 - Month 9; n=17 | -0.5 (2.70)
  CO2 content/Bicarb; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  CO2 content/Bicarb; Visit 6 - Month 12; n=15 | -0.9 (1.44)
  CO2 content/Bicarb; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  CO2 content/Bicarb; Visit 7-(Month 16); n=14 | -0.1 (2.59)
  CO2 content/Bicarb; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  CO2 content/Bicarb; Visit 8 - (Month 20); n=12 | -0.8 (1.96)
  CO2 content/Bicarb; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  CO2 content/Bicarb; Visit 9 - (Month 24); n=11 | -1.5 (2.58)
  CO2 content/Bicarb; Visit 10-(Month 28); n=9: number analyzed (Participants) | 9
  CO2 content/Bicarb; Visit 10-(Month 28); n=9 | -1.8 (1.39)
  CO2 content/Bicarb; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  CO2 content/Bicarb; Visit 11-(Month 32); n=9 | 2.4 (1.94)
  CO2 content/Bicarb; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  CO2 content/Bicarb; Visit 12-(Month 36); n=4 | -1.5 (1.91)
  CO2content/Bicarb;Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  CO2content/Bicarb;Study Conclusion/Withdrawal;n=27 | -1.0 (2.72)
  CO2 content/Bicarb; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  CO2 content/Bicarb; Follow-Up Visit; n=4 | 0.8 (2.36)
  Chloride; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Chloride; Visit 1-Day 1; n=28 | -0.4 (2.97)
  Chloride; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Chloride; Visit 2 - Month 1; n=27 | -0.2 (3.32)
  Chloride; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Chloride; Visit 3 - Month 3; n=24 | -0.2 (2.91)
  Chloride; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Chloride; Visit 4 - Month 6; n=19 | -0.3 (2.89)
  Chloride; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Chloride; Visit 5 - Month 9; n=17 | 0.1 (3.22)
  Chloride; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Chloride; Visit 6 - Month 12; n=15 | 0.6 (3.54)
  Chloride; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Chloride; Visit 7-(Month 16); n=14 | 0.7 (3.73)
  Chloride; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Chloride; Visit 8 - (Month 20); n=12 | 1.3 (3.70)
  Chloride; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Chloride; Visit 9 - (Month 24); n=11 | 1.0 (3.32)
  Chloride; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Chloride; Visit 10-(Month 28); n=10 | 0.9 (3.87)
  Chloride; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Chloride; Visit 11-(Month 32); n=9 | 1.3 (5.32)
  Chloride; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Chloride; Visit 12-(Month 36); n=4 | -1.5 (3.87)
  Chloride; StudyConclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Chloride; StudyConclusion/Withdrawal;n=27 | -0.4 (3.67)
  Chloride; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Chloride; Follow-Up Visit; n=4 | -0.8 (2.22)
  Glucose; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Glucose; Visit 1-Day 1; n=28 | -0.42 (1.458)
  Glucose; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Glucose; Visit 2 - Month 1; n=27 | 0.13 (1.554)
  Glucose; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Glucose; Visit 3 - Month 3; n=24 | 0.12 (1.426)
  Glucose; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Glucose; Visit 4 - Month 6; n=19 | 0.55 (1.094)
  Glucose; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Glucose; Visit 5 - Month 9; n=17 | 0.32 (1.709)
  Glucose; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Glucose; Visit 6 - Month 12; n=15 | 0.05 (1.477)
  Glucose; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Glucose; Visit 7-(Month 16); n=14 | 1.97 (6.817)
  Glucose; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Glucose; Visit 8 - (Month 20); n=12 | 0.08 (1.298)
  Glucose; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Glucose; Visit 9 - (Month 24); n=11 | 0.49 (1.713)
  Glucose; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Glucose; Visit 10-(Month 28); n=10 | 1.14 (2.303)
  Glucose; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Glucose; Visit 11-(Month 32); n=9 | 1.13 (0.892)
  Glucose; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Glucose; Visit 12-(Month 36); n=4 | 1.75 (2.533)
  Glucose; StudyConclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Glucose; StudyConclusion/Withdrawal;n=27 | 0.72 (2.312)
  Glucose; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Glucose; Follow-Up Visit; n=4 | -0.30 (1.152)
  Magnesium; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Magnesium; Visit 1-Day 1; n=28 | -0.004 (0.0522)
  Magnesium; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Magnesium; Visit 2 - Month 1; n=27 | -0.017 (0.0716)
  Magnesium; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Magnesium; Visit 3 - Month 3; n=24 | -0.019 (0.0733)
  Magnesium; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Magnesium; Visit 4 - Month 6; n=19 | -0.016 (0.0565)
  Magnesium; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Magnesium; Visit 5 - Month 9; n=17 | 0.006 (0.0662)
  Magnesium; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Magnesium; Visit 6 - Month 12; n=15 | 0.027 (0.0640)
  Magnesium; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Magnesium; Visit 7-(Month 16); n=14 | 0.041 (0.0434)
  Magnesium; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Magnesium; Visit 8 - (Month 20); n=12 | 0.040 (0.0628)
  Magnesium; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Magnesium; Visit 9 - (Month 24); n=11 | 0.035 (0.0520)
  Magnesium; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Magnesium; Visit 10-(Month 28); n=10 | 0.058 (0.0692)
  Magnesium; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Magnesium; Visit 11-(Month 32); n=9 | 0.050 (0.0585)
  Magnesium; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Magnesium; Visit 12-(Month 36); n=4 | 0.020 (0.0606)
  Magnesium; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Magnesium; Study Conclusion/Withdrawal;n=27 | 0.016 (0.0582)
  Magnesium; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Magnesium; Follow-Up Visit; n=4 | 0.053 (0.1424)
  Potassium; Visit 1-Day 1; n=27: number analyzed (Participants) | 27
  Potassium; Visit 1-Day 1; n=27 | 0.01 (0.277)
  Potassium; Visit 2 - Month 1; n=26: number analyzed (Participants) | 26
  Potassium; Visit 2 - Month 1; n=26 | -0.05 (0.258)
  Potassium; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Potassium; Visit 3 - Month 3; n=24 | 0.00 (0.227)
  Potassium; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Potassium; Visit 4 - Month 6; n=19 | 0.07 (0.341)
  Potassium; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Potassium; Visit 5 - Month 9; n=17 | 0.01 (0.398)
  Potassium; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Potassium; Visit 6 - Month 12; n=15 | 0.10 (0.321)
  Potassium; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Potassium; Visit 7-(Month 16); n=14 | 0.06 (0.247)
  Potassium; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Potassium; Visit 8 - (Month 20); n=12 | 0.09 (0.215)
  Potassium; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Potassium; Visit 9 - (Month 24); n=11 | 0.08 (0.264)
  Potassium; Visit 10-(Month 28); n=9: number analyzed (Participants) | 9
  Potassium; Visit 10-(Month 28); n=9 | 0.21 (0.318)
  Potassium; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Potassium; Visit 11-(Month 32); n=9 | -0.02 (0.367)
  Potassium; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Potassium; Visit 12-(Month 36); n=4 | 0.18 (0.222)
  Potassium; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Potassium; Study Conclusion/Withdrawal;n=27 | -0.02 (0.275)
  Potassium; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Potassium; Follow-Up Visit; n=4 | 0.20 (0.163)
  Sodium; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Sodium; Visit 1-Day 1; n=28 | -0.9 (3.37)
  Sodium; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Sodium; Visit 2 - Month 1; n=27 | -0.3 (3.48)
  Sodium; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Sodium; Visit 3 - Month 3; n=24 | 0.8 (3.00)
  Sodium; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Sodium; Visit 4 - Month 6; n=19 | -0.3 (2.79)
  Sodium; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Sodium; Visit 5 - Month 9; n=17 | 0.7 (2.52)
  Sodium; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Sodium; Visit 6 - Month 12; n=15 | 0.7 (3.58)
  Sodium; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Sodium; Visit 7-(Month 16); n=14 | 0.2 (4.21)
  Sodium; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Sodium; Visit 8 - (Month 20); n=12 | 0.8 (4.13)
  Sodium; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Sodium; Visit 9 - (Month 24); n=11 | 1.1 (2.07)
  Sodium; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Sodium; Visit 10-(Month 28); n=10 | 1.3 (3.53)
  Sodium; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Sodium; Visit 11-(Month 32); n=9 | 1.2 (4.74)
  Sodium; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Sodium; Visit 12-(Month 36); n=4 | -2.0 (4.76)
  Sodium; StudyConclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Sodium; StudyConclusion/Withdrawal;n=27 | 0.2 (3.14)
  Sodium; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Sodium; Follow-Up Visit; n=4 | 0.5 (2.08)
  Urea/BUN; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Urea/BUN; Visit 1-Day 1; n=28 | 0.14 (1.176)
  Urea/BUN; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Urea/BUN; Visit 2 - Month 1; n=27 | 0.36 (1.239)
  Urea/BUN; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Urea/BUN; Visit 3 - Month 3; n=24 | 0.46 (1.353)
  Urea/BUN; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Urea/BUN; Visit 4 - Month 6; n=19 | 0.37 (1.180)
  Urea/BUN; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Urea/BUN; Visit 5 - Month 9; n=17 | 0.62 (0.884)
  Urea/BUN; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Urea/BUN; Visit 6 - Month 12; n=15 | 0.51 (0.877)
  Urea/BUN; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Urea/BUN; Visit 7-(Month 16); n=14 | 0.25 (1.260)
  Urea/BUN; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Urea/BUN; Visit 8 - (Month 20); n=12 | 0.91 (1.372)
  Urea/BUN; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Urea/BUN; Visit 9 - (Month 24); n=11 | 0.46 (1.016)
  Urea/BUN; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Urea/BUN; Visit 10-(Month 28); n=10 | 0.39 (1.325)
  Urea/BUN; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Urea/BUN; Visit 11-(Month 32); n=9 | 0.77 (1.578)
  Urea/BUN; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Urea/BUN; Visit 12-(Month 36); n=4 | 1.90 (1.971)
  Urea/BUN; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Urea/BUN; Study Conclusion/Withdrawal;n=27 | 0.18 (1.409)
  Urea/BUN; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Urea/BUN; Follow-Up Visit; n=4 | 0.25 (1.287)

17. Primary Outcome: Change From Baseline in Creatinine, Direct Bilirubin, Total Bilirubin, and Uric Acid
Description: Blood samples were collected from participants to evaluate change from Baseline in creatinine, direct bilirubin, total bilirubin, and uric acid. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Micromoles per liter (µmol/L)
  Creatinine; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Creatinine; Visit 1-Day 1; n=28 | -2.18 (5.860)
  Creatinine; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Creatinine; Visit 2 - Month 1; n=27 | -0.79 (6.450)
  Creatinine; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Creatinine; Visit 3 - Month 3; n=24 | -0.35 (5.360)
  Creatinine; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Creatinine; Visit 4 - Month 6; n=19 | -1.39 (6.575)
  Creatinine; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Creatinine; Visit 5 - Month 9; n=17 | 0.32 (4.770)
  Creatinine; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Creatinine; Visit 6 - Month 12; n=15 | 0.61 (4.837)
  Creatinine; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Creatinine; Visit 7-(Month 16); n=14 | -0.94 (6.951)
  Creatinine; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Creatinine; Visit 8 - (Month 20); n=12 | -0.05 (5.970)
  Creatinine; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Creatinine; Visit 9 - (Month 24); n=11 | -0.15 (5.095)
  Creatinine; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Creatinine; Visit 10-(Month 28); n=10 | 4.31 (8.665)
  Creatinine; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Creatinine; Visit 11-(Month 32); n=9 | -3.30 (4.268)
  Creatinine; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Creatinine; Visit 12-(Month 36); n=4 | -2.73 (11.099)
  Creatinine; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Creatinine; Study Conclusion/Withdrawal;n=27 | -0.08 (5.467)
  Creatinine; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Creatinine; Follow-Up Visit; n=4 | 4.30 (20.628)
  Direct Bilirubin; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Direct Bilirubin; Visit 1-Day 1; n=28 | -0.2 (0.67)
  Direct Bilirubin; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Direct Bilirubin; Visit 2 - Month 1; n=27 | 0.0 (0.65)
  Direct Bilirubin; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Direct Bilirubin; Visit 3 - Month 3; n=24 | 0.0 (0.46)
  Direct Bilirubin; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Direct Bilirubin; Visit 4 - Month 6; n=19 | 0.0 (0.58)
  Direct Bilirubin; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Direct Bilirubin; Visit 5 - Month 9; n=17 | -0.2 (0.64)
  Direct Bilirubin; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Direct Bilirubin; Visit 6 - Month 12; n=15 | -0.1 (0.35)
  Direct Bilirubin; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Direct Bilirubin; Visit 7-(Month 16); n=14 | -0.1 (0.53)
  Direct Bilirubin; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Direct Bilirubin; Visit 8 - (Month 20); n=12 | -0.1 (0.51)
  Direct Bilirubin; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Direct Bilirubin; Visit 9 - (Month 24); n=11 | -0.2 (0.75)
  Direct Bilirubin; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Direct Bilirubin; Visit 10-(Month 28); n=10 | -0.1 (0.32)
  Direct Bilirubin; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Direct Bilirubin; Visit 11-(Month 32); n=9 | -0.2 (0.44)
  Direct Bilirubin; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Direct Bilirubin; Visit 12-(Month 36); n=4 | 0.0 (0.82)
  Direct Bilirubin; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Direct Bilirubin; Study Conclusion/Withdrawal;n=27 | 0.0 (0.59)
  Direct Bilirubin; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Direct Bilirubin; Follow-Up Visit; n=4 | 0.3 (1.26)
  Total Bilirubin; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Total Bilirubin; Visit 1-Day 1; n=28 | 3.0 (2.57)
  Total Bilirubin; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Total Bilirubin; Visit 2 - Month 1; n=27 | 3.7 (2.69)
  Total Bilirubin; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Total Bilirubin; Visit 3 - Month 3; n=24 | 3.8 (2.14)
  Total Bilirubin; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Total Bilirubin; Visit 4 - Month 6; n=19 | 3.7 (2.87)
  Total Bilirubin; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Total Bilirubin; Visit 5 - Month 9; n=17 | 2.8 (1.85)
  Total Bilirubin; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Total Bilirubin; Visit 6 - Month 12; n=15 | 3.1 (3.03)
  Total Bilirubin; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Total Bilirubin; Visit 7-(Month 16); n=14 | 3.5 (1.65)
  Total Bilirubin; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Total Bilirubin; Visit 8 - (Month 20); n=12 | 2.8 (1.90)
  Total Bilirubin; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Total Bilirubin; Visit 9 - (Month 24); n=11 | 2.7 (1.95)
  Total Bilirubin; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Total Bilirubin; Visit 10-(Month 28); n=10 | 3.0 (2.11)
  Total Bilirubin; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Total Bilirubin; Visit 11-(Month 32); n=9 | 2.6 (1.51)
  Total Bilirubin; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Total Bilirubin; Visit 12-(Month 36); n=4 | 4.5 (2.65)
  Total Bilirubin; Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Total Bilirubin; Study Conclusion/Withdrawal;n=27 | 2.9 (2.83)
  Total Bilirubin; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Total Bilirubin; Follow-Up Visit; n=4 | 2.3 (4.99)
  Uric acid; Visit 1-Day 1; n=28: number analyzed (Participants) | 28
  Uric acid; Visit 1-Day 1; n=28 | -0.6 (31.72)
  Uric acid; Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Uric acid; Visit 2 - Month 1; n=27 | 6.3 (33.86)
  Uric acid; Visit 3 - Month 3; n=24: number analyzed (Participants) | 24
  Uric acid; Visit 3 - Month 3; n=24 | -5.8 (31.63)
  Uric acid; Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Uric acid; Visit 4 - Month 6; n=19 | 0.3 (32.18)
  Uric acid; Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Uric acid; Visit 5 - Month 9; n=17 | 4.3 (25.30)
  Uric acid; Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Uric acid; Visit 6 - Month 12; n=15 | -5.5 (38.81)
  Uric acid; Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Uric acid; Visit 7-(Month 16); n=14 | -15.0 (51.93)
  Uric acid; Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Uric acid; Visit 8 - (Month 20); n=12 | -10.5 (45.12)
  Uric acid; Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Uric acid; Visit 9 - (Month 24); n=11 | 8.6 (51.81)
  Uric acid; Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Uric acid; Visit 10-(Month 28); n=10 | 6.3 (64.91)
  Uric acid; Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Uric acid; Visit 11-(Month 32); n=9 | -5.2 (66.94)
  Uric acid; Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Uric acid; Visit 12-(Month 36); n=4 | -30.3 (46.50)
  Uric acid; Study Conclusion/Withdrawal;n=26: number analyzed (Participants) | 26
  Uric acid; Study Conclusion/Withdrawal;n=26 | 9.7 (46.87)
  Uric acid; Follow-Up Visit; n=4: number analyzed (Participants) | 4
  Uric acid; Follow-Up Visit; n=4 | 15.8 (62.74)

18. Primary Outcome: Change From Baseline in Urine Albumin/Creatinine Ratio
Description: Urine samples were collected from participants to evaluate change from Baseline in urine albumin/creatinine ratio. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated. NA indicates data was not available as standard deviation could not be calculated for single participant.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Ratio
  Visit 1-Day 1; n=22: number analyzed (Participants) | 22
  Visit 1-Day 1; n=22 | -0.05 (1.603)
  Visit 2 - Month 1; n=19: number analyzed (Participants) | 19
  Visit 2 - Month 1; n=19 | 0.16 (0.932)
  Visit 3 - Month 3; n=18: number analyzed (Participants) | 18
  Visit 3 - Month 3; n=18 | 1.51 (5.755)
  Visit 4 - Month 6; n=14: number analyzed (Participants) | 14
  Visit 4 - Month 6; n=14 | -0.32 (1.342)
  Visit 5 - Month 9; n=12: number analyzed (Participants) | 12
  Visit 5 - Month 9; n=12 | -0.26 (1.006)
  Visit 6 - Month 12; n=10: number analyzed (Participants) | 10
  Visit 6 - Month 12; n=10 | 9.80 (31.071)
  Visit 7-(Month 16); n=8: number analyzed (Participants) | 8
  Visit 7-(Month 16); n=8 | 0.69 (1.733)
  Visit 8 - (Month 20); n=7: number analyzed (Participants) | 7
  Visit 8 - (Month 20); n=7 | -0.24 (0.547)
  Visit 9 - (Month 24); n=7: number analyzed (Participants) | 7
  Visit 9 - (Month 24); n=7 | -0.34 (2.070)
  Visit 10-(Month 28); n=6: number analyzed (Participants) | 6
  Visit 10-(Month 28); n=6 | 0.38 (1.450)
  Visit 11-(Month 32); n=6: number analyzed (Participants) | 6
  Visit 11-(Month 32); n=6 | 0.87 (1.519)
  Visit 12-(Month 36); n=1: number analyzed (Participants) | 1
  Visit 12-(Month 36); n=1 | 0.80 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Study Conclusion/Withdrawal;n=17: number analyzed (Participants) | 17
  Study Conclusion/Withdrawal;n=17 | 0.51 (1.715)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 3.30 (7.044)

19. Primary Outcome: Number of Participants With Abnormal Urinalysis Values (Categorical Data)
Description: Urine samples were collected from participants to analyze presence of abnormal urinalysis parameters including glucose, ketones, RBC, WBC, occult blood and protein. Abnormal urinalysis values have been presented for all parameters. Only those participants with data available at specific time points were analyzed (represented by n= X in the category titles).
Time Frame: Up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  Visit 1 Day1, Glucose, 4+or 2 or more g/dL,n=30 | 2
  Visit 1 Day 1, RBC, 1-3,n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 1-3,n=29 | 4
  Visit 1 Day 1, RBC, 3-5, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 3-5, n=29 | 4
  Visit 1 Day 1, RBC, 5-10, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 5-10, n=29 | 6
  Visit 1 Day 1, RBC, 10-15, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 10-15, n=29 | 1
  Visit 1 Day 1, RBC, 15-25, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 15-25, n=29 | 6
  Visit 1 Day 1, RBC, 25-50, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 25-50, n=29 | 2
  Visit 1 Day 1, RBC, 50-100, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, RBC, 50-100, n=29 | 1
  Visit 1 Day 1, WBC,1-3, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, WBC,1-3, n=29 | 3
  Visit 1 Day 1, WBC,3-5, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, WBC,3-5, n=29 | 1
  Visit 1 Day 1, WBC,5-10, n=29: number analyzed (Participants) | 29
  Visit 1 Day 1, WBC,5-10, n=29 | 2
  Visit 1 Day 1, Occult Blood,1+, n=30 | 1
  Visit 1 Day 1, Occult Blood,4+, n=30 | 1
  Visit 1 Day 1, protein, 1+, n=30 | 5
  Visit 2 Month 1, Glucose,1+ or 1/4 g/dL, n=28: number analyzed (Participants) | 28
  Visit 2 Month 1, Glucose,1+ or 1/4 g/dL, n=28 | 1
  Visit 2 Month 1, Glucose,4+or 2 or more g/dL,n=28: number analyzed (Participants) | 28
  Visit 2 Month 1, Glucose,4+or 2 or more g/dL,n=28 | 1
  Visit 2 Month 1, Ketone 1+, n=28: number analyzed (Participants) | 28
  Visit 2 Month 1, Ketone 1+, n=28 | 1
  Visit 2 Month 1, RBC, 1-3, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 1-3, n=27 | 7
  Visit 2 Month 1, RBC, 3-5, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 3-5, n=27 | 4
  Visit 2 Month 1, RBC, 5-10, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 5-10, n=27 | 4
  Visit 2 Month 1, RBC, 10-15, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 10-15, n=27 | 4
  Visit 2 Month 1, RBC, 15-25, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 15-25, n=27 | 1
  Visit 2 Month 1, RBC, 50-100, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, RBC, 50-100, n=27 | 1
  Visit 2 Month 1,WBC,1-3, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1,WBC,1-3, n=27 | 5
  Visit 2 Month 1, WBC,3-5, n=27: number analyzed (Participants) | 27
  Visit 2 Month 1, WBC,3-5, n=27 | 1
  Visit 2 Month 1, Occult Blood,1+, n=28: number analyzed (Participants) | 28
  Visit 2 Month 1, Occult Blood,1+, n=28 | 1
  Visit 2 Month 1, protein, 1+, n=28: number analyzed (Participants) | 28
  Visit 2 Month 1, protein, 1+, n=28 | 5
  Visit 3 Month 3, Ketones,1+, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, Ketones,1+, n=26 | 1
  Visit 3 Month 3, RBC, 1-3, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 1-3, n=26 | 5
  Visit 3 Month 3, RBC, 3-5, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 3-5, n=26 | 3
  Visit 3 Month 3, RBC, 5-10, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 5-10, n=26 | 6
  Visit 3 Month 3, RBC, 10-15, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 10-15, n=26 | 3
  Visit 3 Month 3, RBC, 15-25, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 15-25, n=26 | 2
  Visit 3 Month 3, RBC, 25-50, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC, 25-50, n=26 | 2
  Visit 3 Month 3, RBC,innumerable, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, RBC,innumerable, n=26 | 1
  Visit 3 Month 3, WBC,1-3, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, WBC,1-3, n=26 | 4
  Visit 3 Month 3, WBC,15-25, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, WBC,15-25, n=26 | 3
  Visit 3 Month 3, WBC,innumerable, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, WBC,innumerable, n=26 | 1
  Visit 3 Month 3, Occult Blood,1+, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, Occult Blood,1+, n=26 | 3
  Visit 3 Month 3, Occult Blood,4+, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, Occult Blood,4+, n=26 | 1
  Visit 3 Month 3, protein, 1+, n=26: number analyzed (Participants) | 26
  Visit 3 Month 3, protein, 1+, n=26 | 6
  Visit 4 Month 6, Glucose,3+ or 1 g/dL, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, Glucose,3+ or 1 g/dL, n=19 | 2
  Visit 4 Month 6, RBC, 1-3, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 1-3, n=19 | 5
  Visit 4 Month 6, RBC, 3-5, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 3-5, n=19 | 3
  Visit 4 Month 6, RBC, 5-10, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 5-10, n=19 | 3
  Visit 4 Month 6 RBC, 10-15,n=19: number analyzed (Participants) | 19
  Visit 4 Month 6 RBC, 10-15,n=19 | 1
  Visit 4 Month 6, RBC, 15-25, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 15-25, n=19 | 2
  Visit 4 Month 6, RBC, 25-50, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 25-50, n=19 | 1
  Visit 4 Month 6, RBC, 50-100, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, RBC, 50-100, n=19 | 1
  Visit 4 Month 6, WBC,1-3, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, WBC,1-3, n=19 | 1
  Visit 4 Month 6, WBC,3-5, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, WBC,3-5, n=19 | 1
  Visit 4 Month 6, Occult Blood,1+, n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, Occult Blood,1+, n=19 | 2
  Visit 4 Month 6, protein, 1+,n=19: number analyzed (Participants) | 19
  Visit 4 Month 6, protein, 1+,n=19 | 3
  Visit 5 Month 9, Glucose,2+ or 1/2 g/dL, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, Glucose,2+ or 1/2 g/dL, n=17 | 1
  Visit 5 Month 9, Glucose,3+ or 1 g/dL, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, Glucose,3+ or 1 g/dL, n=17 | 1
  Visit 5 Month 9, RBC, 1-3, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 1-3, n=17 | 1
  Visit 5 Month 9, RBC, 3-5, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 3-5, n=17 | 5
  Visit 5 Month 9, RBC, 5-10, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 5-10, n=17 | 3
  Visit 5 Month 9, RBC, 10-15, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 10-15, n=17 | 3
  Visit 5 Month 9, RBC, 15-25, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 15-25, n=17 | 1
  Visit 5 Month 9, RBC, 25-50, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, 25-50, n=17 | 1
  Visit 5 Month 9, RBC, innumerable, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, RBC, innumerable, n=17 | 1
  Visit 5 Month 9, WBC,1-3, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, WBC,1-3, n=17 | 4
  Visit 5 Month 9, WBC,15-25, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, WBC,15-25, n=17 | 1
  Visit 5 Month 9, WBC, innumerable, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, WBC, innumerable, n=17 | 1
  Visit 5 Month 9,Occult Blood,1+, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9,Occult Blood,1+, n=17 | 1
  Visit 5 Month 9, Occult Blood,4+, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, Occult Blood,4+, n=17 | 2
  Visit 5 Month 9, protein, 1+, n=17: number analyzed (Participants) | 17
  Visit 5 Month 9, protein, 1+, n=17 | 1
  Visit 6 Month 12, RBC, 1-3, n= 15: number analyzed (Participants) | 15
  Visit 6 Month 12, RBC, 1-3, n= 15 | 4
  Visit 6 Month 12, RBC, 3-5, n= 15: number analyzed (Participants) | 15
  Visit 6 Month 12, RBC, 3-5, n= 15 | 3
  Visit 6 Month 12, RBC, 5-10, n= 15: number analyzed (Participants) | 15
  Visit 6 Month 12, RBC, 5-10, n= 15 | 5
  Visit 6 Month 12, RBC, 10-15, n= 15: number analyzed (Participants) | 15
  Visit 6 Month 12, RBC, 10-15, n= 15 | 2
  Visit 6 Month 12, RBC, 15-25, n= 15: number analyzed (Participants) | 15
  Visit 6 Month 12, RBC, 15-25, n= 15 | 1
  Visit 6, Month 12, WBC, 1-3, n= 15: number analyzed (Participants) | 15
  Visit 6, Month 12, WBC, 1-3, n= 15 | 5
  Visit 6, Month 12, WBC, 3-5, n= 15: number analyzed (Participants) | 15
  Visit 6, Month 12, WBC, 3-5, n= 15 | 2
  Visit 6, Month 12, Occult blood, 1+, n= 15: number analyzed (Participants) | 15
  Visit 6, Month 12, Occult blood, 1+, n= 15 | 4
  Visit 6, Month 12, Protein, 1+, n= 15: number analyzed (Participants) | 15
  Visit 6, Month 12, Protein, 1+, n= 15 | 2
  Visit 6, Month 12, Protein, 2+, n= 15: number analyzed (Participants) | 15
  Visit 6, Month 12, Protein, 2+, n= 15 | 1
  Visit 7,Month16,Glucose, 4+ or 2 or more g/dL,n=14: number analyzed (Participants) | 14
  Visit 7,Month16,Glucose, 4+ or 2 or more g/dL,n=14 | 1
  Visit 7, Month 16, Ketone, 1+, n= 14: number analyzed (Participants) | 14
  Visit 7, Month 16, Ketone, 1+, n= 14 | 1
  Visit 7, Month 16, RBC, 1-3, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, RBC, 1-3, n= 13 | 2
  Visit 7, Month 16, RBC, 3-5, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, RBC, 3-5, n= 13 | 2
  Visit 7, Month 16, RBC, 5-10, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, RBC, 5-10, n= 13 | 3
  Visit 7, Month 16, RBC, 10-15, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, RBC, 10-15, n= 13 | 2
  Visit 7, Month 16, RBC, 25-50, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, RBC, 25-50, n= 13 | 2
  Visit 7, Month 16, WBC, 1-3, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, WBC, 1-3, n= 13 | 2
  Visit 7, Month 16, WBC, 3-5, n= 13: number analyzed (Participants) | 13
  Visit 7, Month 16, WBC, 3-5, n= 13 | 1
  Visit 7, Month 16, Occult blood, 1+, n= 14: number analyzed (Participants) | 14
  Visit 7, Month 16, Occult blood, 1+, n= 14 | 1
  Visit 7, Month 16, Occult blood, 4+, n= 14: number analyzed (Participants) | 14
  Visit 7, Month 16, Occult blood, 4+, n= 14 | 1
  Visit 7, Month 16, Protein, 1+, n= 14: number analyzed (Participants) | 14
  Visit 7, Month 16, Protein, 1+, n= 14 | 3
  Visit 8, Month 20, RBC, 1-3, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, RBC, 1-3, n= 12 | 3
  Visit 8, Month 20, RBC, 3-5, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, RBC, 3-5, n= 12 | 2
  Visit 8, Month 20, RBC, 10-15, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, RBC, 10-15, n= 12 | 2
  Visit 8, Month 20, RBC, 15-25, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, RBC, 15-25, n= 12 | 1
  Visit 8, Month 20, RBC, 25-50, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, RBC, 25-50, n= 12 | 1
  Visit 8, Month 20, WBC, 1-3, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, WBC, 1-3, n= 12 | 2
  Visit 8, Month 20, WBC, 3-5, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, WBC, 3-5, n= 12 | 1
  Visit 8, Month 20, Occult blood, 1+, n= 12: number analyzed (Participants) | 12
  Visit 8, Month 20, Occult blood, 1+, n= 12 | 2
  Visit 9,Month24,Glucose,4+ or 2 or more g/dL,n=11: number analyzed (Participants) | 11
  Visit 9,Month24,Glucose,4+ or 2 or more g/dL,n=11 | 1
  Visit 9, Month 24, RBC, 1-3, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, RBC, 1-3, n= 11 | 3
  Visit 9, Month 24, RBC, 3-5, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, RBC, 3-5, n= 11 | 1
  Visit 9, Month 24, RBC, 5-10, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, RBC, 5-10, n= 11 | 2
  Visit 9, Month 24, RBC, 10-15, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, RBC, 10-15, n= 11 | 1
  Visit 9, Month 24, RBC, 50-100, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, RBC, 50-100, n= 11 | 1
  Visit 9, Month 24, WBC, 3-5, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, WBC, 3-5, n= 11 | 1
  Visit 9, Month 24, WBC, Innumerable, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, WBC, Innumerable, n= 11 | 1
  Visit 9, Month 24, Occult blood, 1+, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, Occult blood, 1+, n= 11 | 1
  Visit 9, Month 24, Occult blood, 4+, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, Occult blood, 4+, n= 11 | 2
  Visit 9, Month 24, Protein, 1+, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, Protein, 1+, n= 11 | 1
  Visit 9, Month 24, Protein, 2+, n= 11: number analyzed (Participants) | 11
  Visit 9, Month 24, Protein, 2+, n= 11 | 1
  Visit 10,Month28,Glucose,4+ or 2 or more g/dL,n=10: number analyzed (Participants) | 10
  Visit 10,Month28,Glucose,4+ or 2 or more g/dL,n=10 | 1
  Visit 10, Month 28, RBC, 1-3, n= 9: number analyzed (Participants) | 9
  Visit 10, Month 28, RBC, 1-3, n= 9 | 2
  Visit 10, Month 28, RBC, 3-5, n= 9: number analyzed (Participants) | 9
  Visit 10, Month 28, RBC, 3-5, n= 9 | 2
  Visit 10, Month 28, RBC, 5-10, n= 9: number analyzed (Participants) | 9
  Visit 10, Month 28, RBC, 5-10, n= 9 | 2
  Visit 10, Month 28, RBC, 25-50, n= 9: number analyzed (Participants) | 9
  Visit 10, Month 28, RBC, 25-50, n= 9 | 1
  Visit 10, Month 28, WBC, 1-3, n= 9: number analyzed (Participants) | 9
  Visit 10, Month 28, WBC, 1-3, n= 9 | 1
  Visit 10, Month 28, Occult blood, 1+, n= 10: number analyzed (Participants) | 10
  Visit 10, Month 28, Occult blood, 1+, n= 10 | 1
  Visit 10, Month 28, Protein, 1+, n= 10: number analyzed (Participants) | 10
  Visit 10, Month 28, Protein, 1+, n= 10 | 2
  Visit 11,Month 32,Glucose,4+ or 2 or more g/dL,n=9: number analyzed (Participants) | 9
  Visit 11,Month 32,Glucose,4+ or 2 or more g/dL,n=9 | 1
  Visit 11, Month 32, RBC, 3-5, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, RBC, 3-5, n= 9 | 1
  Visit 11, Month 32, RBC, 5-10, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, RBC, 5-10, n= 9 | 2
  Visit 11, Month 32, RBC, 10-15, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, RBC, 10-15, n= 9 | 2
  Visit 11, Month 32, RBC, 25-50, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, RBC, 25-50, n= 9 | 1
  Visit 11, Month 32, RBC, 50-100, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, RBC, 50-100, n= 9 | 1
  Visit 11, Month 32, WBC, 1-3, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, WBC, 1-3, n= 9 | 1
  Visit 11, Month 32, WBC, 10-15, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, WBC, 10-15, n= 9 | 1
  Visit 11, Month 32, WBC, innumerable, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, WBC, innumerable, n= 9 | 1
  Visit 11, Month 32, Occult blood, 1+, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, Occult blood, 1+, n= 9 | 1
  Visit 11, Month 32, Occult blood, 2+, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, Occult blood, 2+, n= 9 | 1
  Visit 11, Month 32, Occult blood, 4+, n= 9: number analyzed (Participants) | 9
  Visit 11, Month 32, Occult blood, 4+, n= 9 | 1
  Visit 12,Month 36,Glucose,4+ or 2 or more g/dL,n=4: number analyzed (Participants) | 4
  Visit 12,Month 36,Glucose,4+ or 2 or more g/dL,n=4 | 1
  Visit 12, Month 36, RBC, 3-5, n= 4: number analyzed (Participants) | 4
  Visit 12, Month 36, RBC, 3-5, n= 4 | 2
  Visit 12, Month 36, RBC, 5-10, n= 4: number analyzed (Participants) | 4
  Visit 12, Month 36, RBC, 5-10, n= 4 | 1
  Visit 12, Month 36, Occult blood, 1+, n= 4: number analyzed (Participants) | 4
  Visit 12, Month 36, Occult blood, 1+, n= 4 | 1
  Study conclusion/Withdrawal,Glucose,3+or1g/dL,n=28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal,Glucose,3+or1g/dL,n=28 | 1
  Study conclusion/Withdrawal,Glucose,4+or2g/dL,n=28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal,Glucose,4+or2g/dL,n=28 | 2
  Study conclusion/Withdrawal, Ketones, trace, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Ketones, trace, n= 28 | 1
  Study conclusion/Withdrawal, RBC, 1-3, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 1-3, n= 28 | 5
  Study conclusion/Withdrawal, RBC, 3-5, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 3-5, n= 28 | 2
  Study conclusion/Withdrawal, RBC, 5-10, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 5-10, n= 28 | 7
  Study conclusion/Withdrawal, RBC, 10-15, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 10-15, n= 28 | 4
  Study conclusion/Withdrawal, RBC, 15-25, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 15-25, n= 28 | 2
  Study conclusion/Withdrawal, RBC, 25-50, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, RBC, 25-50, n= 28 | 2
  Study conclusion/Withdrawal, WBC, 1-3, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, WBC, 1-3, n= 28 | 4
  Study conclusion/Withdrawal, WBC, 3-5, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, WBC, 3-5, n= 28 | 2
  Study conclusion/Withdrawal, WBC, 5-10, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, WBC, 5-10, n= 28 | 1
  Study conclusion/Withdrawal, WBC 10-15, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, WBC 10-15, n= 28 | 1
  Study conclusion/Withdrawal, WBC 15-25, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, WBC 15-25, n= 28 | 1
  Study conclusion/Withdrawal, Occult blood,1+ n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Occult blood,1+ n= 28 | 2
  Study conclusion/Withdrawal, Occult blood,2+ n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Occult blood,2+ n= 28 | 1
  Study conclusion/Withdrawal, Occult blood,4+ n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Occult blood,4+ n= 28 | 2
  Study conclusion/Withdrawal, Protein, trace, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Protein, trace, n= 28 | 1
  Study conclusion/Withdrawal, Protein, 1+, n= 28: number analyzed (Participants) | 28
  Study conclusion/Withdrawal, Protein, 1+, n= 28 | 5
  Follow up, Ketones, trace, n= 5: number analyzed (Participants) | 5
  Follow up, Ketones, trace, n= 5 | 1
  Follow up, RBC, 1-3, n= 5: number analyzed (Participants) | 5
  Follow up, RBC, 1-3, n= 5 | 1
  Follow up, RBC, 5-10, n= 5: number analyzed (Participants) | 5
  Follow up, RBC, 5-10, n= 5 | 2
  Follow up, WBC, 1-3, n= 5: number analyzed (Participants) | 5
  Follow up, WBC, 1-3, n= 5 | 3
  Follow up, WBC, 10-15, n= 5: number analyzed (Participants) | 5
  Follow up, WBC, 10-15, n= 5 | 1
  Follow up, Protein, 1+, n= 5: number analyzed (Participants) | 5
  Follow up, Protein, 1+, n= 5 | 1

20. Primary Outcome: Specific Gravity of Urine at Indicated Time Points
Description: Urine samples were collected to analyze specific gravity of urine. Specific gravity, is a measure of urine concentration and is measured using a chemical test. Specific gravity measurements provide a comparison of the amount of substances dissolved in urine as compared to pure water. If there were no solutes present, the specific gravity of urine would be 1.000 the same as pure water. Specific gravity between 1.002 and 1.035 could be considered as normal. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilograms per meter^3 (Kg/m^3)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Kilograms per meter^3 (Kg/m^3)
  Visit 1-Day 1; n=30 | 1.0160 (0.00423)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | 1.0157 (0.00522)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | 1.0187 (0.00437)
  Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Visit 4 - Month 6; n=19 | 1.0161 (0.00542)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | 1.0153 (0.00413)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 1.0157 (0.00458)
  Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Visit 7-(Month 16); n=14 | 1.0146 (0.00414)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | 1.0158 (0.00359)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | 1.0145 (0.00350)
  Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10-(Month 28); n=10 | 1.0140 (0.00459)
  Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Visit 11-(Month 32); n=9 | 1.0139 (0.00486)
  Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Visit 12-(Month 36); n=4 | 1.0150 (0.00408)
  Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Study Conclusion/Withdrawal;n=28 | 1.0166 (0.00409)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 1.0198 (0.00476)

21. Primary Outcome: Potential of Hydrogen (pH) of Urine at Indicated Time Points
Description: Urine Samples were collected to analyze pH. pH is a measure of hydrogen ion concentration and used to determine the acidity or alkalinity of urine. pH scale ranges from 0 to 14. A neutral pH is 7.0. The higher number indicates the more basic (alkaline) nature of urine and lower the number indicates the more acidic urine. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Scores on a scale
  Visit 1-Day 1; n=30 | 6.68 (0.771)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | 6.48 (0.659)
  Visit 3 - Month 3; n=26: number analyzed (Participants) | 26
  Visit 3 - Month 3; n=26 | 6.35 (0.784)
  Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Visit 4 - Month 6; n=19 | 6.39 (0.756)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | 6.74 (0.640)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 6.40 (0.828)
  Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Visit 7-(Month 16); n=14 | 6.54 (0.746)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | 6.71 (0.620)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | 6.86 (1.051)
  Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10-(Month 28); n=10 | 6.80 (0.919)
  Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Visit 11-(Month 32); n=9 | 6.78 (0.667)
  Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Visit 12-(Month 36); n=4 | 6.88 (0.250)
  Study Conclusion/Withdrawal;n=28: number analyzed (Participants) | 28
  Study Conclusion/Withdrawal;n=28 | 6.52 (0.687)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 6.10 (0.548)

22. Primary Outcome: Change From Baseline in Urine Creatinine Concentration
Description: Urine samples were collected from participants to evaluate change from Baseline in Urine creatinine concentration. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RTG IR
Number analyzed (Participants) | 30
µmol/L
  Visit 1-Day 1; n=30 | -1803.3 (6012.94)
  Visit 2 - Month 1; n=27: number analyzed (Participants) | 27
  Visit 2 - Month 1; n=27 | -1725.9 (6632.88)
  Visit 3 - Month 3; n=25: number analyzed (Participants) | 25
  Visit 3 - Month 3; n=25 | -508.0 (6155.28)
  Visit 4 - Month 6; n=19: number analyzed (Participants) | 19
  Visit 4 - Month 6; n=19 | -94.7 (7902.92)
  Visit 5 - Month 9; n=17: number analyzed (Participants) | 17
  Visit 5 - Month 9; n=17 | -58.8 (6676.18)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | -286.7 (3000.21)
  Visit 7-(Month 16); n=14: number analyzed (Participants) | 14
  Visit 7-(Month 16); n=14 | -235.7 (3996.27)
  Visit 8 - (Month 20); n=12: number analyzed (Participants) | 12
  Visit 8 - (Month 20); n=12 | -341.7 (7648.46)
  Visit 9 - (Month 24); n=11: number analyzed (Participants) | 11
  Visit 9 - (Month 24); n=11 | -81.8 (5230.07)
  Visit 10-(Month 28); n=10: number analyzed (Participants) | 10
  Visit 10-(Month 28); n=10 | 4940.0 (9857.11)
  Visit 11-(Month 32); n=9: number analyzed (Participants) | 9
  Visit 11-(Month 32); n=9 | 2944.4 (6495.98)
  Visit 12-(Month 36); n=3: number analyzed (Participants) | 3
  Visit 12-(Month 36); n=3 | 1000.0 (11887.39)
  Study Conclusion/Withdrawal;n=27: number analyzed (Participants) | 27
  Study Conclusion/Withdrawal;n=27 | -1781.5 (5805.11)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 7100.0 (4959.33)

23. Primary Outcome: Change From Baseline in American Urological Association (AUA) Symptom Scale Scores
Description: The effect of RTG on bladder function was assessed using AUA symptom index. It is a 7-item Likert-scored scale with seven questions, each with six potential responses. Responses to each of 7 questions were scored from 0 (no symptom at all) to 5 (almost always symptoms present) which were summmed to get total possible score ranging from 0 to 35 with higher scores indicating worse symptom severity. The total score for all questions was classified as mild (0-7), moderate (8-19) or severe (>19). Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Retigabine IR
Number analyzed (Participants) | 30
Scores on a scale
  Visit 1-Day 1; n=29: number analyzed (Participants) | 29
  Visit 1-Day 1; n=29 | -0.5 (2.68)
  Visit 2-Month 1; n=28: number analyzed (Participants) | 28
  Visit 2-Month 1; n=28 | 0.3 (2.37)
  Visit 3 - Month 3; n=25: number analyzed (Participants) | 25
  Visit 3 - Month 3; n=25 | -0.3 (2.41)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | -0.7 (1.58)
  Visit 7-(Month 16); n=1: number analyzed (Participants) | 1
  Visit 7-(Month 16); n=1 | -2.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Visit 9 - (Month 24); n=10: number analyzed (Participants) | 10
  Visit 9 - (Month 24); n=10 | -0.1 (5.20)
  Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Visit 12-(Month 36); n=4 | 3.0 (5.48)
  Visit 13 (Month 40); n=1: number analyzed (Participants) | 1
  Visit 13 (Month 40); n=1 | 0.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Study Conclusion/Withdrawal;n=29: number analyzed (Participants) | 29
  Study Conclusion/Withdrawal;n=29 | 1.1 (4.45)
  Follow-Up Visit; n=5: number analyzed (Participants) | 5
  Follow-Up Visit; n=5 | 1.2 (3.56)

24. Primary Outcome: Change From Baseline in Post-void Residual (PVR) Bladder Ultrasound Volumes
Description: The PVR bladder ultrasound was used to assess the effects of RTG on bladder function. Baseline was defined as the last assessment of that endpoint in parent study RTG114855 taken prior to the first active treatment with RTG IR. Change from Baseline was defined as post-Baseline value minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles). Mean and SD were calculated.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Milliliter (mL)
  Visit 1-Day 1; n=29: number analyzed (Participants) | 29
  Visit 1-Day 1; n=29 | -3.4 (36.38)
  Visit 2 - Month 1; n=28: number analyzed (Participants) | 28
  Visit 2 - Month 1; n=28 | 9.2 (24.66)
  Visit 3 - Month 3; n=25: number analyzed (Participants) | 25
  Visit 3 - Month 3; n=25 | 2.0 (39.72)
  Visit 6 - Month 12; n=15: number analyzed (Participants) | 15
  Visit 6 - Month 12; n=15 | 1.7 (30.67)
  Visit 7-(Month 16); n=1: number analyzed (Participants) | 1
  Visit 7-(Month 16); n=1 | -8.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Visit 9 - (Month 24); n=10: number analyzed (Participants) | 10
  Visit 9 - (Month 24); n=10 | -8.2 (36.79)
  Visit 12-(Month 36); n=4: number analyzed (Participants) | 4
  Visit 12-(Month 36); n=4 | -13.1 (31.50)
  Visit 13 (Month 40); n=1: number analyzed (Participants) | 1
  Visit 13 (Month 40); n=1 | 35.0 (NA) — NA indicates data was not available as standard deviation could not be calculated for single participant.
  Study Conclusion/Withdrawal;n=29: number analyzed (Participants) | 29
  Study Conclusion/Withdrawal;n=29 | -1.7 (31.01)
  Follow-Up Visit; n=3: number analyzed (Participants) | 3
  Follow-Up Visit; n=3 | -22.0 (53.70)

25. Primary Outcome: Number of Participants With Suicidal Ideation or Behavior During Treatment Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Number of participants with suicidal ideation or behavior during treatment were assessed using the C-SSRS score scale. It is a brief questionnaire designed to assess severity and change in suicidality by integrating both behavior and ideation using a semi-structured interview to probe participant responses. It consists of an assessment of suicidal ideation (ranging from "desire to be dead" to "active suicidal ideation with specific plan and intent") and an assessment of suicidal behavior (ranging from "preparatory acts or behavior" to "completed suicide").
Time Frame: Up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  Suicidal ideation | 1
  Suicidal behavior | 0

26. Primary Outcome: Number of Participants Who Discontinued From RTG
Description: The number of participants who discontinued from RTG treatment has been presented.
Time Frame: Up to 4 years
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Participants
  Day 0 | 0
  Day 3 | 1
  Day 17 | 1
  Day 62 | 1
  Day 66 | 1
  Day 98 | 1
  Day 111 | 1
  Day 126 | 1
  Day 163 | 1
  Day 168 | 2
  Day 169 | 1
  Day 229 | 1
  Day 240 | 1
  Day 287 | 1
  Day 339 | 1
  Day 413 | 1
  Day 498 | 1
  Day 559 | 1
  Day 650 | 1
  Day 781 | 1
  Day 852 | 1
  Day 927 | 1
  Day 930 | 0
  Day 943 | 0
  Day 1007 | 1
  Day 1008 | 1
  Day 1098 | 0
  Day 1169 | 0
  Day 1233 | 0

27. Primary Outcome: Percentage of Participants With Retinal Pigmentary Abnormalities
Description: Percentage of participants with abnormal findings after eye examination were evaluated. Abnormalities detected on-treatment in study RTG114873 were presented. Retinal pigmentary abnormalities included abnormalities in the macula, peripheral retina and unspecified location.
Time Frame: Up to 4 years
Population: Safety Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | RTG IR
Number analyzed (Participants) | 22
Percentage of participants | 18

28. Primary Outcome: Percentage of Participants With Pigmentation of Non-retinal Ocular Tissues
Description: Percentage of participants with abnormal findings after eye examination were evaluated. Abnormalities detected on-treatment in study RTG114873 were presented. Pigmentation of non-retinal ocular tissues included pigmentation of the sclera and/or conjunctiva, cornea, iris and lens.
Time Frame: Up to 4 years
Population: Safety Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | RTG IR
Number analyzed (Participants) | 22
Percentage of participants | 32

29. Primary Outcome: Percentage of Participants With Dermatologist-confirmed Abnormal Discoloration
Description: Percentage of participants with abnormal findings after skin examination (including the skin around the eyes and the eyelids, lips, nails, or mucosa) were evaluated.
Time Frame: Up to 4 years
Population: Safety Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | RTG IR
Number analyzed (Participants) | 25
Percentage of participants | 0

30. Primary Outcome: Percentage of Participants With a Clinically Significant Decrease in Visual Acuity From Initial Examination
Description: Percentage of participants with a clinically significant decrease in visual acuity from initial examination were evaluated. Only abnormalities occurring on-treatment in study RTG114873 were presented.
Time Frame: Up to 4 years
Population: Safety Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | RTG IR
Number analyzed (Participants) | 19
Percentage of participants | 16

31. Primary Outcome: Percentage of Participants With Decrease in Confrontational Visual Field From Initial Examination
Description: Percentage of participants with decrease in confrontational visual field from initial examination were evaluated. Only abnormalities occurring on-treatment in study RTG114873 were presented.
Time Frame: Up to 4 years
Population: Safety Population. Only those participants with data available at specific time point were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | RTG IR
Number analyzed (Participants) | 19
Percentage of participants | 21

32. Primary Outcome: Percentage of Responders to POS Frequency
Description: A responder was defined as a participant experiencing a >=50 percent reduction in 28 day total POS frequency from Baseline. A responder rate was calculated overall and based on duration of exposure. As this was an OLE study, Baseline was defined by the parent study Baseline period. Percentage of responders were evaluated from study RTG114873 Day 1 through the last dosing day, excluding the Taper Phase.
Time Frame: Up to 4 years
Population: Safety Population
Measure: Number; unit: Percentage of responders
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Percentage of responders | 23

33. Primary Outcome: Percent Change From Baseline in 28-day Total POS Frequency
Description: The 28-day total POS frequency was calculated as the number of total POS reported during the treatment phase, divided by the number of applicable days in the treatment phase, then multiplying this ratio by 28. In this formula, innumerable seizures were counted as 10 seizures and status epilepticus was counted as 1 seizure. As this was an OLE study, Baseline was defined by the parent study Baseline period. The percent change from Baseline was calculated as the 28-day total POS on-treatment frequency (during dosing in this study, not including the taper phase) minus the Baseline 28-day total POS frequency, with this difference being divided by the Baseline 28-day partial seizure rate, and the resulting quantity multiplied by 100. It was calculated as overall and by duration of exposure. Mean and SD were presented.
Time Frame: Baseline and up to 4 years
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | RTG IR
Number analyzed (Participants) | 30
Percent change | -29.37 (58.363)

34. Primary Outcome: Number of Participants With Resolution of Abnormal Eye Pigmentation After Discontinuation of RTG
Description: The ophthalmologist/retina specialist determined the presence or absence of retinal and non-retinal ocular abnormalities. Retinal abnormalities included abnormalities in the macula and/or the peripheral retina. This analysis was performed on the All SFUCP Subjects population which comprised of all participants who enter the SFUCP.
Time Frame: Up to 1.4 years
Population: All SFUCP Subjects
Measure: Count of Participants; unit: Participants
Groups:
- RTG in SFUCP: Participants who withdraw from the Open-Label Treatment Phase (i.e., discontinue RTG IR including any dose taper), and who were found to have retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP which was the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR.
Arm/Group | RTG in SFUCP
Number analyzed (Participants) | 4
Participants
  Retinal pigmentary abnormality | 0
  Non-retinal ocular pigmentary abnormality | 0

35. Primary Outcome: Number of Participants With Resolution of Dermatologist-confirmed Abnormal Discoloration After Discontinuation of RTG
Description: The skin examination included assessment of the skin around the eyes and the eye lids, lips, nails, and mucosa. Participants who enter the SFUCP who had on-treatment finding(s) of abnormal discoloration of skin, lips, nails or mucosa confirmed by a dermatologist, underwent assessments performed by a dermatologist at 6-monthly intervals.
Time Frame: Up to 1.4 years
Population: All SFUCP Subjects
Measure: Count of Participants; unit: Participants
Arm/Group | RTG in SFUCP
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (non-SAEs) were collected from the start of the study treatment up to 4 years.
Description: AEs and SAEs were collected in "Safety Population" for RTG IR arm and in "All SFUCP Subjects Population" for RTG in SFUCP arm.
Groups:
- RTG in SFUCP: Participants who withdraw from the Open-Label Treatment Phase and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or abnormal discoloration of nails, lips, skin or mucosa were followed-up in SFUCP which was the final reporting phase of the study. During SFUCP, participants underwent six monthly comprehensive eye examinations and/or dermatological assessments. Participants were followed-up until the discoloration /pigmentation either resolves or stabilizes, as defined by no change over two consecutive six monthly assessments over at least 12 months after discontinuation of RTG IR.
Arm/Group | RTG IR | RTG in SFUCP
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/4
Serious Adverse Events (participants affected / at risk) | 5/30 | 0/4
Other Adverse Events (participants affected / at risk) | 23/30 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTG IR (N=30) | RTG in SFUCP (N=4)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0
Endophthalmitis (Infections and infestations) | 1 (1) | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0
Postictal state (Nervous system disorders) | 1 (2) | 0
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0
Dizziness (Nervous system disorders) | 1 (1) | 0
Headache (Nervous system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RTG IR (N=30) | RTG in SFUCP (N=4)
Retinal pigmentation (Eye disorders) | 2 (2) | 0
Vision blurred (Eye disorders) | 2 (2) | 0
Fatigue (General disorders) | 2 (2) | 0
Asthenia (General disorders) | 3 (3) | 0
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0
Nasopharyngitis (Infections and infestations) | 3 (3) | 0
Memory impairment (Nervous system disorders) | 3 (3) | 0
Headache (Nervous system disorders) | 4 (4) | 0
Somnolence (Nervous system disorders) | 9 (10) | 0
Dizziness (Nervous system disorders) | 11 (16) | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.